Mason W. Freeman

| Protocol THR-14 | 42-C-418: Statistical Analysis Plan | Research" |
|---|---|---|
| TIOOOOI IMEE IT | The Title Statistical Additions of the | <u> ಎರಡಿ ಕ್ರೀಟ್ ಕ್ರವಾಗಿ ಕ್ರಿಟ್ ಕ್ರೀಟ್ ಕ್ರಾಲೀಕ ಕ್ರೀಟ್ ಚಾರ್ ಗಾರ್ಗೌಸ್ಟ್ ಕ್ರೀಟ್ ಕ್ರಟ್ ಕ್ರಟ್ ಕ್ರೀಟ್ ಕ್ರಟ್ ಕ</u> |
| Signature Page | | |
| | , | |
| I confirm that I ha | eve reviewed this document and agree with the content. | * |
| | agion with the continue | en e |
| Theracos, Inc. | | |
| Trice | | |
| Signature: | 11 1. 31 0 | 11 500 7 -16 |
| | Yuan-Di Halvorsen | Nov. 28, 2011 |
| | | Date |
| | Senior Clinical Research Project Leader | |
| | A. Tark | |
| Signature: | 7101101 | Ha) 198 2011 |
| | Monica Tettamanti | Date |
| | Clinical Trial Manager | |
| | / | |
| Signature: | Mason W. Freuer | Nov 28 2011 |
| | Mason Freeman | Nov 28 2011 |
| | Medical Monitor | Date |
| | MACGICAL MICHIGA | A STATE OF THE STA |
| INC Research, 1 | LLC | |
| Signature: | No Allen | 29 M0020 11 |
| • | Vicky Pan | 29 N0020 1 |
| | Project Biostatistician | |
| Signature: | Naver Xmonden - Way | 79 Non- 7011 |
| · · · | Karen Snowdon-Way, MS | 29 Nov- 2011<br>Date |
| | Reviewing Biostatistician | Date |
| | A / | |
| Pion man | Mohlankarlas | 2011/2020 |
| Signature: | | 29 NOV2011 |
| | Ašhley Kesler | Date |
| | Lead Statistical Togrammer | |
| | $\mathcal{L}$ | |
| Signature: | May / Lon. | 29 No 2011 |
| | Nancy Chau | Date |
| | Project Leader | |
| | <b>₩</b> | • |

Final - 22November 2011

CONFIDENTIAL




## STATISTICAL ANALYSIS PLAN

INC RESEARCH PROJECT: 021815

AUTHOR: Vicky Pan

INC RESEARCH PROJECT

LEADER:

DATE OF ISSUE: 22 November 2011

SAP VERSION: Final

SPONSOR: Theracos, Inc.

STUDY TITLE: Efficacy and safety of EGT0001442 compared

Nancy Chau

with placebo in patients with type 2 diabetes mellitus inadequately controlled by diet and exercise and up to one oral anti-diabetes agent

PROTOCOL NUMBER: Protocol THR-1442-C-418

PROTOCOL VERSION/DATE: Amendment 3 (12 September 2011)

### Confidentiality Statement

The following confidential information is the property of Theracos, Inc. As long as the information contained in this document has not been published, it may only be used when permission has been obtained from Theracos



Date

## Protocol THR-1442-C-418: Statistical Analysis Plan

## Signature Page

Signature:

Nancy Chau

Project Leader

I confirm that I have reviewed this document and agree with the content.

| Theracos, Inc. | | |
|-----------------------------|-----------------------------------------|------|
| Signature: | | |
| | Yuan-Di Halvorsen | Date |
| | Senior Clinical Research Project Leader | |
| Signature: | | |
| | Monica Tettamanti | Date |
| | Clinical Trial Manager | |
| Signature: | | |
| | Mason Freeman | Date |
| | Medical Monitor | |
| INC Research, L. Signature: | LC | |
| | Vicky Pan | Date |
| | Project Biostatistician | |
| Signature: | | |
| | Karen Snowdon-Way, MS | Date |
| | Reviewing Biostatistician | |
| Signature: | | |
| | Ashley Kesler | Date |
| | Lead Statistical Programmer | |



## **Table of Contents**

| st of Abb | reviations and Definitions of Terms | 5 |
|---|---|---|
| Study | Objectives | 7 |
| | • • | |
| _ | | |
| | • | |
| | v | |
| 3.6.1 | • | |
| 3.6.2 | Final Analysis | 14 |
| | - | |
| 5.1 Pr | otocol Deviations | 15 |
| 5.3.1 | Last Observation Carried Forward. | 16 |
| 5.3.2 | | |
| 5.4 As | ssessment Windows | 17 |
| 5.4.1 | Study Day | 17 |
| 5.4.2 | Visit Slotting Algorithm | 17 |
| 5.4.3 | Multiple Evaluations | 18 |
| 5.5 Si | te Pooling | 19 |
| Demog | graphics, Baseline Characteristics, and Medications | 19 |
| | <u> </u> | |
| | Genera 1.1 Pu 1.2 Re 1.1 Pu 1.2 Re 1.2 Study 2.1 Pr 2.2 Se 1.3 Study 3.1 Br 3.2 Su 3.3 As 3.4 Bl 3.5 Sa 3.6 PI 3.6.1 3.6.2 Analys 4.1 Sa 4.2 Fu 4.3 Pe 4.4 De Genera 5.1 Pr 5.2 M 5.3 M 5.3.1 5.3.2 5.4 As 5.4.1 5.4.2 5.4.3 5.5 Si Demog 6.1 Su 6.2 De 6.3 M | General Considerations 1.1 Purpose 1.2 Responsibilities Study Objectives 2.1 Primary Objective 2.2 Secondary Objectives Study Design 3.1 Brief Description 3.2 Subject Selection 3.3 Assessment Schedule 3.4 Blinding, Randomization, and Bias 3.5 Sample Size Justification 3.6 PLANNED ANALYSES 3.6.1 Week 24 Analysis 3.6.2 Final Analysis Analysis Sets 4.1 Safety Analysis Set 4.2 Full Analysis Set 4.3 Per Protocol Analysis Set 4.4 Deviations from Assigned Treatment General Consideration for Data Analyses 5.1 Protocol Deviations 5.2 Multiple Comparisons and Multiplicity 5.3 Missing Data Algorithm 5.3.1 Last Observation Carried Forward 5.3.2 Post-rescue Measurements 5.4 Assessment Windows 5.4.1 Study Day 5.4.2 Visit Slotting Algorithm 5.4.3 Multiple Evaluations 5.5 Site Pooling Demographics, Baseline Characteristics, and Medications 6.1 Subject Disposition and Withdrawals 6.2 Demographics and Subject Characteristics at Baseline 6.3 Medical History |



| Protocol THR-1442-C-418: | Statistical Analysis Plan |
|--------------------------|---------------------------|

| 7 Efficacy | |
|---|---|
| <ul><li>7.1 Primary Efficacy Analyses</li><li>7.2 Secondary Efficacy Analyses</li></ul> | |
| 7.2.1 HbA1c Change from Baseline over Time | |
| 7.2.2 FPG Change from Baseline over Time | |
| 7.2.3 Body Weight Change from Baseline over Time | |
| 7.2.4 Blood Pressure Change from Baseline over Time | |
| <ul> <li>7.2.5 Proportion of Subjects who Achieved HbA1c &lt; 7% Response Levels</li> <li>7.3 Exploratory Efficacy Analyses</li> </ul> | 23 |
| 7.3.1 Repeated Measures Analyses | 23 |
| 7.3.2 Analysis of Covariance | 24 |
| 7.3.3 Sensitivity Analyses | 24 |
| 8 Exposure and Compliance 8.1 Extent of Exposure to Study Drug 8.2 Subject Compliance | 25 |
| 9 Safety | |
| 9.1 Adverse Events | |
| 9.1.1 All and Treatment Emergent AEs | 26 |
| 9.1.2 Deaths, Serious AEs, and AEs That Led to Discontinuation | 26 |
| 9.1.3 Adverse Events of Special Interest | |
| 9.2.1 Hematology, Chemistry and Urinalysis | 27 |
| 9.2.2 Drug Screen Results | 28 |
| 9.2.3 Pregnancies | 28 |
| <ul><li>9.2.4 Nuclear Mitotic Apparatus Protein 22 (NMP22) Testing Results</li><li>9.3 Vital Signs and Physical Exams</li></ul> | |
| 9.3.1 Vital Signs | 28 |
| 9.3.2 Physical Exam | |
| 10 Changes in the Conduct of the Study or Planned Analyses | 29 |
| Appendix 1: Table, Figure and Listing Shells | 30 |



# **List of Abbreviations and Definitions of Terms**

| Abbreviation | Definition of Term |
|--------------|----------------------------------------------|
| ADA | American Diabetes Association |
| AE | adverse event |
| AESI | adverse events of special interest |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| ANOVA | analysis of variance |
| AST | aspartate aminotransferase |
| ATC | anatomical/therapeutic/chemical |
| BMI | body mass index |
| BUN | blood urea nitrogen |
| CBC | complete blood count |
| CRF | case report form |
| CVE | cardiovascular event |
| DSMB | data and safety monitoring board |
| ECG | electrocardiogram |
| FAS | full analysis set |
| FPG | fasting plasma glucose |
| HbA1c | glycosylated hemoglobin A1c |
| IWRS | interactive web response system |
| LOCF | last observation carried forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NMP22 | nuclear mitotic apparatus protein 22 |
| OC | observed case |



| PT | preferred term |
|---------|-------------------------------------------|
| RBC | red blood cell |
| SAP | statistical analysis plan |
| SOC | system organ class |
| T2DM | type 2 diabetes mellitus |
| TEAE | treatment emergent adverse event |
| ULN | upper limit of normal |
| WBC | white blood cell |
| WHODRUG | World Health Organization Drug Dictionary |



### 1 General Considerations

## 1.1 Purpose

The purpose of this Statistical Analysis Plan (SAP) is to describe the analyses that will be performed, to ensure that the data listings, summary tables and figures that will be produced and the statistical methodologies that will be used are complete and appropriate to reach valid conclusions regarding the study objectives. In particular, this SAP addresses analyses and reports to be provided using data from the following study:

Clinical Trial Protocol THR-1442-C-418: Efficacy and safety of EGT0001442 compared with placebo in subjects with type 2 diabetes mellitus inadequately controlled by diet and exercise and up to one oral anti-diabetes agent.

## 1.2 Responsibilities

The INC Research Data Management department maintains the clinical database for the trial. The INC Research Biostatistics and Statistical Programming departments will provide data summaries.

# 2 Study Objectives

# 2.1 Primary Objective

The primary objective of this study is to assess the efficacy of EGT0001442 in lowering HbA1c at week 24 compared with placebo.

# 2.2 Secondary Objectives

The secondary objectives of this study are:

- To assess the efficacy of EGT0001442 in lowering FPG at weeks 2 and 24 compared with placebo
- To assess the efficacy of EGT0001442 based on the proportion of subjects who reach the American Diabetes Association (ADA) target HbA1c of <7% in the EGT0001442 group compared with placebo
- To assess the effect of EGT0001442 on systolic and diastolic blood pressure compared with placebo
- To assess the effect of EGT0001442 on body weight compared with placebo
- To assess the change in HbA1c change over time, week 1 to week 96



• To assess the safety of EGT0001442 in patients with T2DM

## 3 Study Design

## 3.1 Brief Description

THR-1442-C-418 is a multinational, 2 arm parallel group, randomized, double-blind placebo-controlled study to compare treatment with once daily EGT0001442, 20 mg capsules to matching placebo in either treatment-naïve type 2 diabetic subjects (i.e. those not taking an anti-hyperglycemic agent for ≥16 weeks prior to study entry) or subjects treated with one oral anti-diabetes drug. The study design consists of a screening period, a 2-week placebo run-in (washout) period, and a 96-week double-blind treatment period. The primary analysis will take place after 24 weeks of double-blind treatment.

In the proposed study, diabetic subjects will be screened within 3 weeks of washout start. At screening visit, subjects who meet all the inclusion criteria, none of the exclusion criteria, and who consent to participate in the study will receive counseling for appropriate diet and exercise. Those who are on an oral anti-diabetic medication will discontinue the medication and receive placebo in this run-in period for  $14 \pm 3$  days. Eligible diabetic subjects who are treatment naïve and who control their hyperglycemia through diet and exercise will also receive placebo and the hyperglycemia will be monitored to ensure that their fasting blood glucose levels remain below 250 mg/dL during this interval of  $14 \pm 3$  days.

After the run-in period, approximately 300 subjects will complete the baseline assessment on day 1, after overnight fasting to confirm their eligibility. The subjects that remain eligible will be randomly assigned in a 1:1 ratio to receive either once daily EGT0001442 in 20 mg capsules or matching placebo, using a computer-generated allocation schedule. Randomization will be stratified by study center and screening HbA1c ( $\geq$ 7 to <8.5% or  $\geq$ 8.5 to  $\leq$ 10%). Each subject will be provided with study drug for 24 weeks, dosing instructions, diet and exercise counseling, and a glycemic control card for recording food and fasting glucose information on the days prior to each clinic visit

Each subject will be instructed to return to the clinic on weeks 2, 6, 12, 18, and 24 for safety monitoring and efficacy assessment including review of adverse events, concomitant medication, vital signs, ECG, physical examination, testing of blood chemistry and hematology laboratory parameters, and a urinalysis.

Subjects who complete the 24-week treatment period will continue receiving the study drug for an additional 72 weeks. Subjects who receive rescue medication due to poor glycemic control will continue to receive approved anti-diabetic medications and standard of care per investigator

Final – 22November2011 



decision, according to current treatment guidelines, during the 72 week follow-on period. In the weeks 25 to 96 treatment period, subjects must return to the clinic on weeks 36, 48, 60, 72, 84, and 96 for continuous safety monitoring and efficacy assessment, including review of HbA1c values, adverse events, concomitant medication, ECG, vital signs, and physical examinations. A follow up exit visit will be conducted one week after the last dose.

The overall study duration from screening until follow-up could last a maximum of 102 weeks for study subjects.

An independent Data and Safety Monitoring Board (DSMB) will monitor overall safety information during the EGT0001442 development program including this study. The safety review activity and potential risk benefit assessments utilized by the DSMB are documented in DSMB charter and a separate DSMB statistical analysis plan.

An independent cardiovascular adjudication committee is established to review cardiovascular events (CVE) occurring during the study, in a blinded fashion. These events include cardiovascular mortality, myocardial infarction, stroke, and hospitalization for acute coronary syndromes, urgent revascularization procedures, and other possible serious cardiovascular events. The adjudicated events will be documented and archived to allow a meta-analysis to be performed to assess if there is any increase in cardiovascular risk to an unacceptable extent at the time of completion of all phase 2 and 3 clinical studies. The evaluation and analysis of adjudicated cardiovascular events will be documented in a separate CVE statistical analysis plan.

This reporting and analysis plan for protocol THR-1442-C-418 will examine several efficacy and safety endpoints at planned analyses time points (described in Section 3.6). Two independent statistical teams from INC Research will analyze data from this study. One team will perform all planned blinded analyses during study conduct, as well as the final end-of-study unblinded analysis (i.e., after all subjects have completed 96 weeks and final follow-up, and the database has been locked.) The second team will perform planned unblinded analyses during the study conduct for continuous safety assessment by the DSMB and interim Week 24 analysis.

## 3.2 Subject Selection

The study population will include approximately 300 subjects diagnosed with T2DM that are inadequately controlled by diet and exercise or by treatment with a single oral anti-diabetes agent and who have an HbA1c level between 7% and 10%. The study will recruit subjects from approximately 35 trial centers in 4 countries.

### 3.3 Assessment Schedule

The study activities at each clinic visit are presented in the following table.

Final – 22November2011 



**Table 1: Schedule of Events** 

| | | ening<br>un-in | | Treati | nent w | eeks 1 | to 24 | | | Treati | nent w | eeks 25 | to 96 | | Follow<br>Up <sup>8</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 |
| Time to Randomization Visit (weeks) <sup>1</sup> | -5 | -2 | 0 | 2 | 6 | 12 | 18 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 1 wk<br>f/u |
| Informed Consent | X | | | | | | | | | | | | | | |
| Screening for I/E criteria | X | X | X | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | |
| Diet & exercise counseling <sup>2</sup> | | X | | | | X | | X | | X | | X | | | |
| Diary & glucometer record review | | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Discontinue anti-diabetic medication | | X | | | | | | | | | | | | | |
| Randomization | | | X | | | | | | | | | | | | |
| Physical exam <sup>3</sup> | X | | | | | X | | X | | X | | X | | X | X |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ECG | X | | X | | | | | X | | | X | | | X | X |
| Dispense study medication | | X | X | | X | X | X | X | X | X | X | X | X | | |
| Blood draw for clinical lab test <sup>4</sup> | X | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis <sup>5</sup> | X | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| NMP22 testing <sup>6</sup> | X | | X | | | | | X | | X | | X | | X | |
| $AE^7$ | | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Con Med | | _ | X | X | X | X | X | X | X | X | X | X | X | X | X |

Screening period may last up to 21 days (V1 to V2), Run-in period is to be 14±3 days (V2 to V3), V3 to V8 window is ±3 days, all other visit windows are the nominal duration from randomization ± 6 days.

Glucose meter will be dispensed at visit 2. Training on using glucometer and recording hyper- or hypoglycemia will be conducted on visit 2.



- A complete physical examination will be performed by the investigator at screening and at the termination visit. An abbreviated physical examination will include body weight and general assessment of the skin, heart, lungs and abdomen. Abbreviated physical examinations will be performed by the investigator at all other time points, unless clinically indicated.
- <sup>4</sup> Blood sample for these lab tests at the designated visit are listed as following. Fasting state must be confirmed.
  - V1: CBC, electrolytes, BUN, creatinine, Lipids (TG, TC, HDL-C), ALT, AST, bilirubin (total and direct), PT, HbA1c, FPG, TSH, Hepatitis Screen (HBsAg, HBcAb, HCV), serum pregnancy for women of childbearing potential
  - V3: CBC, electrolytes, BUN, creatinine, Lipids (TG, TC, HDL-c), ALT, AST, bilirubin (total and direct), HbA1c, FPG
  - V4: CBC, electrolytes, BUN, creatinine, HbA1c, FPG
  - V5: CBC, electrolytes, BUN, creatinine, HbA1c, FPG
  - V6: CBC, electrolytes, BUN, creatinine, Lipids (TG, TC, HDL-c), ALT, AST, bilirubin (total and direct), HbA1c, FPG
  - V7: CBC, electrolytes, BUN, creatinine, HbA1c, FPG
  - V8-V15 and ET: CBC, electrolytes, BUN, creatinine, Lipids (TG, TC, HDL-c), ALT, AST, bilirubin (total and direct), HbA1c, FPG. PT only at V8, and V15 or ET.
- Clean catch sample to be collected at each visit and sent to the central lab. Urine drug screen on screening (visit 1). On-site urine dipstick to be performed at all visits except V2.
- NMP22 testing will be performed at screening (V1), randomization (V3), and at weeks 24 (V8), 48 (V10), 72 (V12), and 96 (V14) or when clinically indicated. For subjects who do not have baseline NMP22 testing following Protocol Amendment 1 (11 April, 2011), NMP22 testing will be performed in the next visit or within 4 weeks after Amendment is approved, whichever comes first.
- Adverse events of special interest are specified to be:
  - Cardio- and cerebro- vascular events.
  - Genitourinary infections
  - Increase in creatinine from baseline by 0.5 mg/dL or more
  - Increase in ALT, AST or bilirubin to >3x ULN
- Visit to be conducted one week after last dose of study drug whether subject early terminates from study or completes V14.



## 3.4 Blinding, Randomization, and Bias

Eligible subjects who complete the  $14 \pm 3$  day run-in period and meet all study inclusion/exclusion requirements will be randomized in a 1:1 ratio to receive EGT0001442 20 mg/day or placebo according to a computer-generated randomization schedule. Subjects will be assigned to treatment groups in sequential order as they qualify for the study, using a centrally located and managed interactive web response system (IWRS). Randomization will be stratified by study center and screening HbA1c ( $\geq 7$  to < 8.5% or  $\geq 8.5$  to 10%). The study will be conducted at multiple investigative sites and will likely involve variable numbers of subjects at each site. Enrollment will be on a competitive basis but each site will be capped at 15% of the total randomized subjects (45 subjects).

The study drug will be blinded to the sponsor, investigators, study coordinators, pharmacists, study subjects, and the cardiovascular adjudication committee members. Upon randomization, each subject will receive a subject randomization number and drug kit(s) assigned to the subject. To maintain blinding of the treatment, the values of the HbA1c after dosing starts will remain blinded to all study personnel and subjects until all subjects have completed the 24 week treatment period. After all subjects have completed the 24 week treatment period, all previous and subsequent HbA1c values will be made available to the sponsor, investigators, study coordinators, pharmacists, and the study subjects for close monitoring of subjects' safety including assessment of providing rescue medication. Subjects' treatment assignment will continue to be held from all study personnel so the remainder of the study can be conducted in a blinded fashion.

If knowledge of the test substance is needed to manage the subject's condition, the investigator will contact the IWRS to obtain the treatment assignment. If unblinding occurs for any reason, the time and reason for unblinding will be recorded on the case report form (CRF) and the sponsor must be notified within 24 hours.

A designated statistician who is not involved with the study operation will hold the treatment code. The unblinded treatment information can be provided to the DSMB to facilitate the evaluation of any clinically important increase in the rate of a serious suspected adverse reaction or to the designated safety contact when the treatment information is required to determine if an expedited safety report must be submitted to regulatory agencies.

The treatment code will be unblinded after all subjects have completed the planned 96 weeks of blinded study treatment and the subsequent follow-up phase, and the clinical database has been locked



The treatment assignment will continue to be withheld from the cardiovascular adjudication committee members at the conclusion of the study until all phase 2 and 3 investigational studies are completed and a meta-analysis to assess cardiovascular risk is conducted.

## 3.5 Sample Size Justification

Approximately 300 subjects will be enrolled and equitably allocated to receive either EGT0001442 20 mg capsules or placebo.

The sample size of 150 subjects per group was calculated based on the following assumptions:

- The mean change from baseline to Week 24 in HbA1c in the active dose group will be approximately -0.4%.
- The placebo group will not experience a substantive mean change in HbA1c from baseline to week 24.
- The standard deviation of this change is the same for both groups and is 1.0%.
- The two groups are independent, the study design is balanced, and the two-sided significance level for the hypothesis is 0.05.

Under the above assumptions, an evaluable sample size of 133 evaluable subjects per treatment arm yields approximately 90% power that EGT0001442 treatment will be found to be significantly different from placebo. A sample size of 150 subjects per treatment arm will be enrolled to account for any subject lost-to-follow-up.

### 3.6 PLANNED ANALYSES

Tests of programming and statistical analyses will commence after data have been collected and are available in the database. This initial testing phase will be performed using dummy treatment codes to maintain the treatment blind.

### 3.6.1 Week 24 Analysis

A limited unblinded analysis will be performed after all subjects have achieved the Week 24 primary efficacy endpoint (at the Week 24 visit), after all subject data up to Week 24 have been cleaned and locked. The purpose of the analysis will be to support management decisions about continuing the EGT0001142 development program. The unblinded results will be provided to a limited number of recipients at Theracos, and will not be made available to any other personnel involved in the study conduct. Subjects will continue to receive their randomized treatment in a blinded manner for the remainder of the planned 96 weeks of treatment and the follow-up phase.

Final – 22November2011 



The Week 24 analysis will be treated as an interim analysis with regard to the blinding and data handling. Since the primary efficacy analysis is conducted once at the Week 24 time point, no multiplicity adjustment will be used for the interim analysis.

### 3.6.2 Final Analysis

After all subjects have completed the planned 96 weeks of blinded study treatment and the subsequent follow-up phase, the final analysis for the clinical study report will be completed. At this time, the database will be frozen, and the treatment codes will be unblinded.

## 4 Analysis Sets

## 4.1 Safety Analysis Set

All subjects who are randomized and administered at least one dose of double-blind study medication will be included in the Safety Analysis Set. The safety analysis set will be used in safety analysis detailed in Section 9. All analyses using the safety analysis set will be analyzed according to treatment received.

## 4.2 Full Analysis Set

The full analysis set (FAS) will include all subjects in the safety analysis set who have a baseline and at least one post-baseline HbA1c measurement. The full analysis set will be used in efficacy analysis detailed in Section 7. All analyses of the full analysis set will be based on randomly assigned treatment.

## 4.3 Per Protocol Analysis Set

The Per Protocol Analysis set will include all subjects in the full analysis set who meet the study inclusion requirements and who have no major protocol deviations that would affect the validity of the efficacy measurements. The definition of major protocol deviations that would result the subject being excluded from the per protocol analysis set is detailed in Section 5.1.

The per protocol analysis set will be used in sensitivity efficacy analyses detailed in Section 7.3.3. All analyses using the per protocol analysis set will be based on randomly assigned treatment.

# 4.4 Deviations from Assigned Treatment

If a subject's actual treatment deviates from the randomly assigned treatment, the extent of the deviation and the type of data being analyzed will be considered in deciding how to assign the subject for analysis.



- If a subject takes the unassigned study medication for only part of the study, the subject will be analyzed based on the randomized treatment assignment for both safety and efficacy.
- If a subject takes the unassigned study medication for the entire study, the subject will be analyzed based on the treatment actually taken for safety analyses. However, the subject will be analyzed according to randomized treatment for efficacy per the intent-to-treat principle.

## 5 General Consideration for Data Analyses

Statistical analyses and summaries of safety and tolerability will be performed using SAS® software version 9.2 or later (SAS Institute, Cary, NC). In all cases, statistical testing and confidence intervals will be two-tailed and significance will be judged at the  $\alpha$ =0.05 level.

### **5.1 Protocol Deviations**

Subject compliance to the protocol will be evaluated prior to unblinding the study and subjects with major protocol deviations will be identified. Specific criteria for what constitutes a major protocol deviation will be determined by the study team. The following criteria will be considered:

- Failure to meet key inclusion/exclusion criteria
- Use of prohibited concomitant medications
- Noncompliance with the study medication dosing schedule

Protocol deviations will be tracked by the clinical team using TrialWatch on an on-going basis and will be listed by subject. A table summary by treatment group and listing of major protocol deviations will be presented by subject for all randomized subjects.

# 5.2 Multiple Comparisons and Multiplicity

There is a single primary endpoint in this study and no correction for multiple comparisons is needed. All other secondary and exploratory analyses which do not qualify for formal statistical testing will not be corrected for multiplicity, and will have results presented with confidence intervals and nominal p-values.

# 5.3 Missing Data Algorithm

Final – 22November 2011 



Imputation of partial or missing dates for the determination of prior/concomitant medication status is addressed in Section 6.4 of this SAP. Imputation of partial or missing dates for the determination of treatment-emergence of adverse events, and handling of missing adverse event data related to event severity or relationship to study drug, are addressed in Section 9.1.

Subjects who discontinue from the study early will not be replaced. For some analyses, the last non-missing observation for a subject may be carried forward (LOCF).

#### 5.3.1 Last Observation Carried Forward

Imputation for missing observations will be applied to selected efficacy endpoints by using the last observation carried forward method. For subjects who withdraw from the study, the last valid observation recorded on treatment (scheduled or unscheduled) will be carried forward to all remaining visits. Also, for subjects in efficacy analyses who had missing observations prior to their last observation on treatment, the closest previous non-missing on-treatment observation will be carried forward to missing visits. If a subject had missing observation(s) immediately after baseline, the baseline observation will not be carried forward and the visit(s) will be left as missing.

In general, the LOCF method will be used for all efficacy endpoints that are evaluated at or before Week 24. Beyond Week 24, all analyses will not impute any missing data; this non-imputation method will be referred to as the observed case (OC). The descriptive summaries of endpoints by study medication group will include the count of missing values at each visit. The detail of which analysis utilizes LOCF algorithm is available in Section 7.

It is expected that 24 weeks of treatment is required to obtain the full treatment effect; shorter treatment periods may result in the observation of only a partial (smaller) treatment effect. Therefore, assuming that subject discontinuation of study drug or early termination from study will occur equally and at random in both treatment groups and in each stratum, this LOCF imputation approach is expected to provide a statistically conservative estimate for the treatment effect.

#### 5.3.2 Post-rescue Measurements

For subjects who are rescued for hyperglycemia, their post-rescue measurements of efficacy parameters will be handled in the same manner as missing values for the efficacy analyses. Post-rescue measurements of efficacy parameters may be included in limited exploratory analyses.

Post-rescue measurements of safety parameters will be included in analyses without any special handling.



#### **5.4** Assessment Windows

### **5.4.1 Study Day**

When study day is used for display or in comparisons the following algorithm will be used:

- study day = date of assessment date of first dose +1, if date of assessment ≥ first dose date
- study day = date of assessment date of first dose, if date of assessment < first dose date.

Note that the date of first dose is Day 1 and the day before the date of first dose is Day -1 (there is no Day 0).

## 5.4.2 Visit Slotting Algorithm

For all safety and efficacy parameters to be summarized or analyzed by visit, data records will be slotted to one of the protocol specified visits using the following algorithm:

- a) Determine the study day for all records using the algorithms from Section 5.4.1
- b) For all records (including unscheduled visit records, early withdrawal records and repeat visit records), use the study day determined above with the slotting intervals in the analysis visit window table below to slot the record to the appropriate analysis visit.

Final – 22November 2011 



**Table 2: Analysis Visit Windows** 

| Scheduled Visit | Target Study Day of Visit | Slotting Intervals |
|---|---|---|
| Week -5 (Screening) | -35 | <=-25 |
| Week -2 | -14 | -24 to -4 days |
| Baseline (Week 0) | 1 | -3 to 1 days |
| Week 2 | 15 | 2 to 29 days |
| Week 6 | 43 | 30 to 64 days |
| Week 12 | 85 | 65 to 106 days |
| Week 18 | 127 | 107 to 148 days |
| Week 24 | 169 | 149 to 211 days |
| Week 36 | 253 | 212 to 295 days |
| Week 48 | 337 | 296 to 379 days |
| Week 60 | 421 | 380 to 463 days |
| Week 72 | 505 | 464 to 547 days |
| Week 84 | 589 | 548 to 631 days |
| Week 96 (End of Treatment | 673 | 632 to (last dose date) |
| Visit)* | | |
| Week 97** | 680 | >Last dose date + 7 days |
| 1 Week Follow-up Visit** | Last dose date + 7 days | >Last dose date + 7 days |

<sup>\*</sup> Week 96 is the end of treatment visit for those subjects completing the study per protocol. For subjects who withdraw early from active treatment, the end of treatment visit will be assigned to an analysis visit based on the visit slotting algorithm using study day.

For parameters which were not scheduled to be collected at all visits, still use the all-inclusive visit intervals defined for all visits (that is, the visit window table above) to slot records. However, if a value is slotted to a visit unscheduled for a parameter, it will not be summarized except for summaries focusing on extreme values such as laboratory shift tables. These records will also be included in data listings.

### **5.4.3** Multiple Evaluations

After all the records have been slotted based on study day, if there are multiple valid records for an assessment within an assigned analysis visit, only one of these records will be used for summary statistics and analyses. The record to be used is determined using the following hierarchy (in decreasing order):

- the record closest to the target visit day
- the record with an original nominal visit that matches the analysis visit

<sup>\*\*</sup> Week 97 is the 1 week post-treatment follow-up visit for those subjects completing the study per protocol. The 1 Week Follow-up Visit is the 1 week post-treatment follow-up visit for those subjects who withdraw early from active treatment.



• the record earliest in time

For missing values prior to Week 24 where the LOCF algorithm is applied, it is always the last valid assessment on treatment carried forward even though this might not be the assessment obtained by the above hierarchy and used in the summaries by visit.

## 5.5 Site Pooling

The study will be conducted at approximately 35 US and international study sites and 4 countries (United States, Mexico, Columbia, and India). Sites will be pooled if appropriate for exploratory efficacy analyses detailed in Section 7.3. Within each country, all sites will be pooled together to form one pooled site, so that a total of 4 pooled sites are available for analyses. At the end of the study, if any single country (such us United States) enrolls significantly more subjects than any other country, a further break-down within that country might be considered as part of the pooling strategy (i.e., regions within United States may be utilized as pooled sites).

# 6 Demographics, Baseline Characteristics, and Medications

## **6.1 Subject Disposition and Withdrawals**

The number of subjects who were randomized and the number of subjects within each analysis set (Safety, Full, Per Protocol) will be summarized for each treatment group. A summary of subjects randomized by country and site will also be provided by treatment group.

Subject status in study participation will be summarized in relation to completion of active treatment through Week 24, and in relation to completion of study. Reasons for early discontinuation of study will be summarized for each treatment group.

Subject disposition data will be listed as well. All disposition summaries will be performed using all randomized subjects. A by-country summary will be provided as well.

The number of subjects who were run-in failures, and the number of subjects who failed to fulfill one or more of the inclusion/exclusion criteria will be tabulated and listed for all run-in failure subjects.

# 6.2 Demographics and Subject Characteristics at Baseline

Demographic data (age, gender, race, ethnicity), baseline characteristics (height, weight, BMI, child bearing potential, baseline HbA1c category) will be summarized.

Final – 22November 2011 



Subject age (years) will be calculated as the full years passed since birth date until the date of informed consent signed:

Age=integer part of [(date of informed consent signed – date of birth + 1) / 365.25].

The BMI will be calculated in kg/m<sup>2</sup>:

 $BMI = body weight [kg] / (height [m])^2$ 

Demographic data and baseline characteristics will be tabulated for each analysis set. Baseline comparability of treatments for demographic and baseline characteristics will be assessed using ANOVA model statistics for continuous variables and chi-square statistics for categorical variables. A by-country summary will be provided using the safety analysis set.

Summary of substance (alcohol, tobacco, and drug) use (both categorical and quantitative) will be produced as well as a by-subject listing. All summaries will be performed using the safety analysis set.

## 6.3 Medical History

The number and percentage of subjects with medical history condition will be reported by treatment group. A summary of duration of diabetes disease history in years will be provided. The duration of diabetes disease history is calculated as the years lapsed between screening visit date and type 2 diabetes diagnosis date. For partial missing diagnosis date, the missing month is imputed as January and the missing day is imputed as the first of the month to calculate duration. All other detailed diabetes medical history will be summarized in total, and by country.

In addition, a by-subject listing for detailed diabetes medical history will be provided, and all other medical history data will be listed. All summaries will be performed using the safety analysis set.

# **6.4 Prior/Concomitant Medications**

Any prior and concomitant medication used during the study will be recorded and coded using World Health Organization Drug Dictionary (WHODRUG) enhanced version June 2011 to obtain a preferred term (PT) and an anatomical/therapeutic/chemical (ATC) level 4 term. Summary of all medications by treatment group, ATC level 4 term and preferred term will be provided.

The date and time of first dose of study drug will be used as cutoff time point for definition of prior and concomitant medication. Prior medications are those started before the first dose of double-blind study drug. Concomitant medications are those taken at any time on or after the

Final – 22November2011 



day of the first dose of double-blind study drug, including those medications that were started prior to randomization but were continued into the double-blind treatment period.

Partial start dates of prior and concomitant medications will be assumed to be the earliest possible date consistent with the partial date. In the case of a missing year, the year will be assumed to be the year part of informed consent date of that subject. In the case of a completely missing start date, the start date will be assumed to be prior to date of the first administration of study drug. Partial stop dates of prior and concomitant medications will be assumed to be the latest possible date consistent with the partial date. In the case of completely missing stop date, medication will be assumed to be ongoing.

All recorded anti-diabetic medications will be included in the medication summaries described above. Those anti-diabetic medications that the investigators indicated as being rescue medications for hyperglycemia will also be summarized separately by treatment group. The number and percent of subject who are rescued for hyperglycemia over time will be tabulated.

All prior and concomitant medications will be listed. All summaries will be performed using the safety analysis set.

## 7 Efficacy

## 7.1 Primary Efficacy Analyses

The primary efficacy endpoint is HbA1c change from baseline at Week 24. The primary hypothesis is that EGT0001442 reduces HbA1c after 24 weeks of treatment when compared to placebo controls. The Week 24 mean change from baseline will be analyzed using a 2 sample t-test between treatment groups. The primary analyses will be performed on the full analysis set using the LOCF algorithm. Subjects who are rescued for hyperglycemia before Week 24 will have their HbA1c recorded at the time of rescue and carried forward for primary analyses. Subjects who discontinue from active treatment due to any reason before Week 24 will also have their last post-baseline HbA1c observation carried forward for the analyses.

# 7.2 Secondary Efficacy Analyses

## 7.2.1 HbA1c Change from Baseline over Time

The continuous secondary efficacy endpoint of HbA1c change from baseline by visit will be analyzed analogous to the primary endpoint using a 2 sample t-test. One analysis will be performed using the LOCF algorithm for all visits, and a separate analysis will be performed using OC algorithm. The OC algorithm analysis will exclude any post-rescue values.

Final – 22November2011 



The pattern of HbA1c over time and change from baseline over time will be evaluated both descriptively using summary statistics and graphically at each scheduled visit during the entire duration of the study, excluding post-rescue measurements. Descriptive summaries will also be provided including post-rescue measurements.

The analyses will be performed on the full analysis set and all data will be listed.

### 7.2.2 FPG Change from Baseline over Time

The continuous secondary efficacy endpoints of FPG change from baseline at Week 2 and Week 24 and FPG change from baseline by visit will be analyzed analogous to the primary endpoint using a 2 sample t-test. One analysis will be performed using the LOCF algorithm for all visits, and a separate analysis will be performed using OC algorithm. The OC algorithm analysis will exclude any post-rescue values.

The pattern of FPG over time and change from baseline over time will be evaluated both descriptively using summary statistics and graphically at each scheduled visit during the entire duration of the study, excluding post-rescue measurements. Descriptive summaries will also be provided including post-rescue measurements.

The analyses will be performed on the full analysis set and all data will be listed.

## 7.2.3 Body Weight Change from Baseline over Time

The continuous secondary efficacy endpoint of body weight change from baseline at Week 2 and Week 24 and body weight change from baseline by visit will be analyzed analogous to the primary endpoint using a 2 sample t-test. One analysis will be performed using the LOCF algorithm for all visits, and a separate analysis will be performed using OC algorithm. The OC algorithm analysis will exclude any post-rescue values.

The pattern of weight over time and change from baseline over time will be evaluated both descriptively using summary statistics and graphically at each scheduled visit during the entire duration of the study, excluding post-rescue measurements. Descriptive summaries will also be provided including post-rescue measurements.

The analysis will be performed on the full analysis set and all data will be listed.

### 7.2.4 Blood Pressure Change from Baseline over Time

The continuous secondary efficacy endpoints of blood pressure (both systolic and diastolic) change from baseline at Week 2 and Week 24 and blood pressure change from baseline by visit will be analyzed analogous to the primary endpoint using a 2 sample t-test. Multiple

Final – 22November2011 



measurements made on the same day will be averaged to measure blood pressure on that day. One analysis will be performed using the LOCF algorithm for all visits, and a separate analysis will be performed using OC algorithm. The OC algorithm analysis will exclude any post-rescue values

The pattern of blood pressure over time and change from baseline over time will be evaluated both descriptively using summary statistics and graphically at each scheduled visit during the entire duration of the study, excluding post-rescue measurements. Descriptive summaries will also be provided including post-rescue measurements.

The analysis will be performed on the full analysis set and all data will be listed.

### 7.2.5 Proportion of Subjects who Achieved HbA1c < 7% Response Levels

The categorical secondary efficacy endpoint of the proportion of subjects achieving HbA1c < 7% response level by visit will be analyzed by treatment comparisons that utilize a chi-square test. One analysis will be performed using the LOCF algorithm for all visits, and a separate analysis will be performed by visit using the OC algorithm. The OC algorithm analysis will exclude any post-rescue values.

The pattern of the response data over time will be evaluated descriptively using summary statistics at each scheduled visit during the entire duration of the study, excluding post-rescue measurements. Descriptive summaries will also be provided including post-rescue measurements.

The analysis will be performed on the full analysis set and all data will be listed.

## 7.3 Exploratory Efficacy Analyses

### 7.3.1 Repeated Measures Analyses

To assess treatment as an effect over time on HbA1c change from baseline, a repeated measures analysis will be performed in supportive of the primary and secondary efficacy analyses. All observed measurements, excluding post-rescue measurements, of change from baseline in HbA1c through Week 96 will be included in the linear mixed effect model as repeated measures. Intercept and slope for time (entered as continuous variable) will be specified as random covariates, which may be simplified as fixed covariates depending on the assessment of the model fit. The PROC MIXED procedure in SAS will be used. The unstructured correlation for repeated HbA1c change from baseline will be specified; if the model fails to converge, an alternative correlation matrix will be specified.



As with HbA1c, repeated measures analyses will also be performed on change from baseline of body weight, systolic blood pressure, diastolic blood pressure, and FPG. A linear effect model will be utilized for each of the change from baseline measures similarly to that being used for HbA1c change from baseline. All analyses will be performed on the full analysis set.

### 7.3.2 Analysis of Covariance

To assess treatment effect adjusted for important covariates on HbA1c change from baseline, an analysis of covariance (ANCOVA) model will be performed in supportive of the primary and secondary efficacy analyses. HbA1c change from baseline by visit will be analyzed using an ANCOVA model with treatment group, site (pooled as necessary), gender (male versus female), race (categorized as white, black, and other non-white), and age (categorized as <65 years, and ≥65 years) as factors and baseline HbA1c as a continuous covariate. One analysis will be performed using the LOCF algorithm for all visits, and a separate analysis will be performed using OC algorithm. The OC algorithm analysis will exclude any post-rescue values.

As with HbA1c, ANCOVA analyses will also be performed on change from baseline of body weight, systolic blood pressure, diastolic blood pressure, and FPG. For each of these endpoint, the ANCOVA model will include treatment group, site (pooled as necessary), gender (male versus female), race (categorized as white, black, and other non-white), age (categorized as <65 years, and ≥65 years), and baseline HbA1c category (≥7 to <8.5% versus ≥8.5 to ≤10%) as factors and corresponding baseline endpoint measures (i.e., baseline FPG for FPG change from baseline ANCOVA mode) as a continuous covariate. All analyses will be performed on the full analysis set.

### 7.3.3 Sensitivity Analyses

When subjects' compliance to the protocol are poor and would affect the validity of the efficacy measurements, sensitivity analyses will be conducted on selected efficacy endpoints by excluding those subjects (i.e., using the per protocol analysis set).

For HbA1c change from baseline by visit, similar analyses of those performed using the full analysis set will be performed using the per protocol analysis set. Both t-test and ANCOVA analyses will be repeated using the LOCF algorithm for all visits. Additionally, the pattern of HbA1c over time and change from baseline over time will be evaluated descriptively using summary statistics at each scheduled visit during the entire duration of the study, excluding post-rescue measurements.

Other efficacy endpoints to be used in sensitivity analyses include FPG change from baseline over time, body weight change from baseline over time, systolic and diastolic blood pressure change from baseline over time, and proportion of subjects achieving HbA1c < 7% response



level over time. The analysis of each of the endpoint will follow the same process described above for HbA1c. All analyses will be performed on the per protocol analysis set.

## 8 Exposure and Compliance

## 8.1 Extent of Exposure to Study Drug

Descriptive summary statistics including the number of subjects, mean, standard deviation, median, minimum, and maximum for the duration of study drug exposure will be presented by treatment group. The duration of study drug exposure is defined as the number of weeks between the date of the first dose and the date of the last dose plus 1 day (that is, exposure in weeks =  $\left[\text{date of last dose - date of first dose} + 1 \text{ day}\right] / 7$ .)

The number and percent of subject who receive at least one dose of double-blind study medication, and the number and percent who complete at least 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, and 96 weeks of treatment will be tabulated.

A by-subject listing of study drug administration will also be presented.

## 8.2 Subject Compliance

Subjects will be given the investigational double-blind drug beginning at Day 1 (Week 0) through Week 96. Investigational product accountability will be done at each study visit after the Week 0 visit through the end-of-treatment visit. Subjects will be instructed to return all unused investigational product at the Week 96 visit in order to perform drug accountability and determine compliance.

The number of administered capsules will be calculated as the number dispensed minus (the number returned plus the number reported as lost/missing and not taken). Treatment compliance will be calculated as total number of administered capsules divided by total number of capsules which should have been taken based on the last completed visit during active treatment period. Treatment compliance will be summarized for all subjects. Summary statistics for treatment compliance percentages, as well as the number and percentage of subjects who are <80%, and ≥80% compliant will be reported for the safety analysis set. Individual subject compliance information will be listed also.

# 9 Safety

All safety summaries and analyses will be performed using the safety analysis set.

Final – 22November2011 



#### 9.1 Adverse Events

### 9.1.1 All and Treatment Emergent AEs

All AEs will be coded using MedDRA version 14.0. A treatment-emergent adverse event (TEAE) is one with a start date on or after the date of the first administration of study drug. Only TEAEs will be included in summary tables. All AEs will be included in listings.

Partial start dates of AE will be assumed to be the earliest possible date consistent with the partial date. In the case of a missing year, the year will be assumed to be the year part of informed consent date of that subject. In the case of a completely missing start date, the start date will be assumed to be prior to date of the first administration of study drug.

In general, AEs will be presented in descending order from the system organ class (SOC) with the highest total incidence (that is, summed across all treatment groups) for any adverse event within the class to the SOC with the lowest total incidence. Within the SOC level, AEs will be presented in descending order from the MedDRA preferred term (PT) with the highest total incidence to the PT with the lowest total incidence. If the total incidence for any two or more PTs within an SOC is equal, the PTs will be presented in alphabetical order. A PT will not be presented if no adverse events occur within the level. At each SOC and PT level of summarization, a subject will be counted once if he/she reports 1 or more events at that level.

A summary of the number and percentage of subjects with TEAEs by severity (mild, moderate, and severe) will be produced. Subjects who experience the same event several times, with different severity will only be counted once according to the maximum severity experienced at each level of summarization. AEs with missing severity will be considered to be severe for the purposes of summarization.

TEAEs will also be summarized in a table by relationship to study drug (related versus not related to study drug). Events reported as not related or unlikely will be categorized as not related; events reported as possible, probable, definite, unknown will be categorized as related. If a relationship to the study drug is missing or unknown, it will be assumed, for the purpose of analyses, to be treatment-related.

A summary of most common TEAEs, defined as any AE on the preferred term level that has an incidence rate >5% among the subjects in either treatment groups, will be produced by treatment.

### 9.1.2 Deaths, Serious AEs, and AEs That Led to Discontinuation

Final – 22November2011 



Serious treatment emergent adverse events will be summarized. Data will be categorized and presented in a manner similar to that described above for the general AE summaries by treatment group. By subject listings of deaths and serious non-fatal AEs will be presented.

A summary of the number and percentage of subjects with TEAEs leading to treatment discontinuation will also be presented by treatment group. A by-subject listing of all AEs leading to treatment discontinuation will be produced.

### 9.1.3 Adverse Events of Special Interest

Categories of adverse events of special interest (AESIs) include:

- Cardiovascular events: myocardial infarction, cerebrovascular stroke, acute coronary syndrome, cardiovascular death, new or exacerbated congestive heart failure, and etc.
- Hypoglycemic events
- Renal and urinary disorders: nocturia, pollakiuria, polyuria, dysuria, and etc.
- Genitourinary infection: cystitis, urethritis, pyelonephritis, balanitis, vulvovaginitis and etc.
- Liver related events.
- Cancer events.
- Bone fracture events.

All AESIs will be identified by appropriate MedDRA preferred term. A by-subject listing of each category of AESI will be produced. Additional information collected for hypoglycemic events including ADA severity and intervention will be tabulated and listed.

### **9.2** Labs

### 9.2.1 Hematology, Chemistry and Urinalysis

Laboratory parameters include the following tests: hematology, chemistry, and urinalysis. Established or generally acknowledged methods, normal ranges, and quality control procedures will be supplied by the local and central laboratory for the study records.

Hematology parameters used in summaries include hematocrit, hemoglobin, platelet count, red blood cell (RBC) count, and white blood cell (WBC) count with differential. Chemistry

Final – 22November2011 



parameters (including lipids) used in summaries include albumin, ALT, AST, blood urea nitrogen, calcium, bicarbonate, chloride, direct bilirubin, glucose, magnesium, phosphorus, potassium, sodium, total bilirubin, total protein, uric acid, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, and ApoB. Urinalysis parameters used in summaries include appearance, bilirubin, color, glucose, ketones, microscopic examination of sediment, nitrites, occult blood, pH, protein, specific gravity, and urobilinogen.

All laboratory parameters will be summarized for each treatment group, at every assessed time point using descriptive statistics and graphical displays of the means and standard deviations over time. In addition, for hematology and chemistry laboratory parameters, changes from baseline in these quantitative tests will be summarized by treatment group and at every assessed post-baseline time point.

Shift tables will be developed by first classifying the subject laboratory results as low, normal, or high in comparison to the applicable laboratory reference range. The number and percentage of subjects with indicated shifts (low, normal, high) in their results from baseline to each post-baseline assessment will be presented for all hematology, chemistry and applicable urinalysis parameters. All laboratory data will be listed.

### 9.2.2 Drug Screen Results

All laboratory data will be listed including urine drug screen and virology results at screening. Such laboratory parameters include HBsAG, HBcAG, HCV Ab, amphetamines, barbiturates, cocaine, metabolites, opiates, benzodiazepines and cannabinoids.

### 9.2.3 Pregnancies

A listing of subject pregnancies confirmed by serum pregnancy test will be provided.

### 9.2.4 Nuclear Mitotic Apparatus Protein 22 (NMP22) Testing Results

NMP22 testing results will be summarized for each treatment group, at every assessed time point, as well as presented in a by-subject listing.

## 9.3 Vital Signs and Physical Exams

### 9.3.1 Vital Signs

The vital sign summary and analysis will be based on the recordings of the variables pulse, temperature and respiration rate. Each vital sign parameter at every assessed time point will be summarized using descriptive statistics and presented graphically. Change from baseline will also be summarized, and all vital sign data will be listed.

### 9.3.2 Physical Exam

Final – 22November2011 



The number and percentage of subjects with normal or abnormal findings in each assessment time point will be reported for each treatment groups and body systems. All physical exam data will be listed.

### **9.4 ECGs**

Each ECG parameter at each assessed time point will be summarized by treatment group using descriptive statistics and presented graphically. Change from baseline will also be summarized. A summary of the number and percentage of subjects on overall ECG interpretation and abnormal findings will be displayed by treatment group.

Additionally, a summary of the number and percent of subjects who experience QT  $\geq$ 450 msec, QT  $\geq$ 480 msec, QT  $\geq$ 500 msec, QTcB  $\geq$ 450 msec, QTcB  $\geq$ 480 msec, QTcB  $\geq$ 500 msec, QTcF  $\geq$ 480 msec, QTcF  $\geq$ 500 msec will be provided,

All ECG data will be listed.

# 10 Changes in the Conduct of the Study or Planned Analyses

Not applicable.

Final – 22November2011 



# Appendix 1: Table, Figure and Listing Shells

# Table, Listing, and Figure Shells

| Table 14.1-1.1.1 Subject Disposition for Run-in Failures (All Enrolled Subjects) | 6 |
|---|---|
| Table 14.1-1.1.2 Subject Disposition for Randomized Subjects (All Randomized Subjects) | 7 |
| Table 14.1-1.1.3 Subject Disposition for Randomized Subjects by Country (All Randomized Subjects) | 9 |
| Table 14.1-1.2 Subjects Randomized by Country and Study Site (All Randomized Subjects) | 10 |
| Table 14.1-1.3 Inclusion/Exclusion Criteria Not Met (All Run-in Failures) | 11 |
| Table 14.1-1.4.1 Demographics and Baseline Characteristics (Safety Analysis Set) | 13 |
| Table 14.1-1.4.2 Demographics and Baseline Characteristics (Full Analysis Set) | 16 |
| Table 14.1-1.4.3 Demographics and Baseline Characteristics (Per Protocol Analysis Set) | 16 |
| Table 14.1-1.4.4 Demographics and Baseline Characteristics by Country (Safety Analysis Set) | 16 |
| Table 14.1-1.5 Substance Use (Safety Analysis Set) | 17 |
| Table 14.1-2.1 Medical History (Safety Analysis Set) | 18 |
| Table 14.1-2.2 Diabetes Disease History (Safety Analysis Set) | 19 |
| Table 14.1-2.3 Diabetes Disease History by Country (Safety Analysis Set) | |
| Table 14.1-3.1 Prior Medications (Safety Analysis Set) | |
| Table 14.1-3.2 Concomitant Medications (Safety Analysis Set) | |
| Table 14.1-3.3 Hyperglycemia Rescue Medications (Safety Analysis Set) | |
| Table 14.1-3.4 Proportion of Subjects with Hyperglycemia Rescue (Safety Analysis Set) | |
| Table 14.1-4.1 Treatment Exposure (Safety Analysis Set) | |
| Table 14.1-4.2 Treatment Compliance (Safety Analysis Set) | |
| Figure 14.2-1.1 Line Graph of Mean (+/- SE) Change from Baseline in HbAlc (%), Excluding Post-Rescue Value | |
| (Full Analysis Set - OC) | 27 |
| Figure 14.2-1.2 Line Graph of Mean (+/- SE) HbA1c (%), Excluding Post-Rescue Values (Full Analysis Set - | 20 |
| OC) | 28 |
| Figure 14.2-2.1 Line Graph of Mean (+/- SE) Change from Baseline in Fasting Plasma Glucose (mmol/L), | 20 |
| Excluding Post-Rescue Values (Full Analysis Set - OC) | 28 |
| | . 28 |
| Figure 14.2-3.1 Line Graph of Mean (+/- SE) Change from Baseline in Weight (kg), Excluding Post-Rescue | . 20 |
| Values (Full Analysis Set - OC) | 29 |
| Figure 14.2-3.2 Line Graph of Mean (+/- SE) Weight (kg), Excluding Post-Rescue Values (Full Analysis Set - | |
| OC) | |
| Figure 14.2-4.1 Line Graph of Mean (+/- SE) Change from Baseline in Systolic Blood Pressure (mmHg), | |
| Excluding Post-Rescue Values (Full Analysis Set - OC) | 29 |
| Figure 14.2-4.2 Line Graph of Mean (+/- SE) Systolic Blood Pressure (mmHg), Excluding Post-Rescue Values | |
| (Full Analysis Set - OC) | 30 |

Protocol: THR-1442-C-418 Page x of y Figure 14.2-5.1 Line Graph of Mean (+/- SE) Change from Baseline in Diastolic Blood Pressure (mmHq), Figure 14.2-5.2 Line Graph of Mean (+/- SE) Diastolic Blood Pressure (mmHq), Excluding Post-Rescue Values Table 14.2-1.1 Analysis of Change from Baseline in HbA1c (%) at Week 24 (Full Analysis Set - LOCF) .......31 Table 14.2-1.3 Analysis of Change from Baseline in HbA1c (%), Excluding Post-Rescue Values (Full Analysis Table 14.2-1.4 Repeated Measures Analysis of Change from Baseline in HbA1c (%) at Week 96, Excluding Post-Table 14.2-2.1 Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L) at Week 24 (Full Table 14.2-2.2 Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L) (Full Analysis Set -LOCF) 38 Table 14.2-2.3 Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L), Excluding Post-rescue Table 14.2-2.4 Repeated Measures Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L) at Table 14.2-2.5 Summary Statistics for Fasting Plasma Glucose (mmol/L) (Full Analysis Set- OC)......40 Table 14.2-2.6 Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L) (Per Protocol Analysis Table 14.2-3.1 Analysis of Change from Baseline in Weight (kg) at Week 24 (Full Analysis Set - LOCF) .......41 Table 14.2-3.2 Analysis of Change from Baseline in Weight (kg) (Full Analysis Set - LOCF) .......41 Table 14.2-3.3 Analysis of Change from Baseline in Weight (kg), Excluding Post-rescue Values (Full Analysis Table 14.2-3.4 Repeated Measures Analysis of Change from Baseline in Weight (kg) at Week 96, Excluding Table 14.2-3.6 Analysis of Change from Baseline in Weight (kg) (Per Protocol Analysis Set - LOCF) .......43 Table 14.2-4.1 Analysis of Change from Baseline in Systolic Blood Pressure (mmHq) at Week 24 (Full Analysis Table 14.2-4.2 Analysis of Change from Baseline in Systolic Blood Pressure (mmHq) (Full Analysis Set -Table 14.2-4.3 Analysis of Change from Baseline in Systolic Blood Pressure (mmHg), Excluding Post-rescue 

| Protocol: THR-1442-C-418 Page x c | of y |
|---|---|
| Table 14.2-4.4 Repeated Measures Analysis of Change from Baseline in Systolic Blood Pressure (mmHg) at We | ek |
| 96, Excluding Post-rescue Values (Full Analysis Set - OC) | |
| Table 14.2-4.5 Summary Statistics for Systolic Blood Pressure (mmHg) (Full Analysis Set- OC) | 46 |
| Table 14.2-4.6 Analysis of Change from Baseline in Systolic Blood Pressure (mmHg) (Per Protocol Analysis | |
| Set - LOCF) | 46 |
| Table 14.2-5.1 Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg) at Week 24 (Full | |
| Analysis Set - LOCF) | 47 |
| Table 14.2-5.2 Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg) (Full Analysis Set - | |
| LOCF) | 47 |
| Table 14.2-5.3 Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg), Excluding Post-rescue | |
| Values (Full Analysis Set- OC) | 48 |
| Table 14.2-5.4 Repeated Measures Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg) at | |
| Week 96, Excluding Post-rescue Values (Full Analysis Set - OC) | |
| Table 14.2-5.5 Summary Statistics for Diastolic Blood Pressure (mmHg) (Full Analysis Set- OC) | |
| Table 14.2-5.6 Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg) (Per Protocol Analysis | |
| Set - LOCF) | |
| Table 14.2-6.1 Analysis of Proportion of Subjects Achieving HbA1c <7% (Full Analysis Set- LOCF)<br>Table 14.2-6.2 Analysis of Proportion of Subjects Achieving HbA1c <7%, Excluding Post-Rescue Values (Ful | |
| | . <u>.</u><br>51 |
| Table 14.2-6.3 Summary Statistics for Proportion of Subjects Achieving HbA1c <7% by Visit (Full Analysis | |
| Set- OC) | |
| Table 14.2-6.4 Analysis of Proportion of Subjects Achieving HbA1c <7% (Per Protocol Analysis Set- LOCF) | |
| Figure 14.3-2.1 Line Graph of Mean (+/- SE) Results for Hematology (Safety Analysis Set) | |
| Figure 14.3-2.2 Line Graph of Mean (+/- SE) Results for Chemistry (Safety Analysis Set) | |
| Figure 14.3-3.1 Line Graph of Mean (+/- SE) Results for Vital Signs (Safety Analysis Set) | |
| Figure 14.3-4.1 Line Graph of Mean (+/- SE) ECG Results (Safety Analysis Set) | |
| Table 14.3-1.1 Overall Summary of Adverse Events (Safety Analysis Set) | |
| Table 14.3-1.2 Treatment Emergent Adverse Events (Safety Analysis Set) | |
| Table 14.3-1.3 Treatment Emergent Adverse Events by Severity (Safety Analysis Set) | |
| Table 14.3-1.4 Treatment Emergent Adverse Events by Relationship to Study Drug (Safety Analysis Set) | |
| Table 14.3-1.5 Most Common Treatment Emergent Adverse Events (Safety Analysis Set) | |
| Table 14.3-1.6 Serious Treatment Emergent Adverse Events (Safety Analysis Set) | |
| Table 14.3-1.7 Treatment Emergent Adverse Events Leading to Treatment Discontinuation (Safety Analysis | |
| Get) | 61 |
| Table 14.3-1.8 Treatment Emergent Hypoglycemic Events by Severity and Intervention (Safety Analysis Set) | |
| Table 14.3-2.1 Change from Baseline in Hematology (Safety Analysis Set) | 63 |
| Table 14.3-2.2 Change from Baseline in Chemistry (Safety Analysis Set) | 64 |

| Protocol: THR-1442-C-418 | Page x of y |
|---|---|
| Table 14.3-2.3 Urinalysis (Safety Analysis Set) | 65 |
| Table 14.3-2.4 Shift in Hematology (Safety Analysis Set) | 66 |
| Table 14.3-2.5 Shift in Chemistry (Safety Analysis Set) | 67 |
| Table 14.3-2.6 Shift in Urinalysis (Safety Analysis Set) | 67 |
| Table 14.3-3.1 Change from Baseline in Vital Signs (Safety Analysis Set) | 68 |
| Table 14.3-4.1 Change from Baseline in ECG Values (Safety Analysis Set) | |
| Table 14.3-4.2 Overall ECG Interpretations and Abnormal Findings (Safety Analysis Set) | 69 |
| Table 14.3-4.3 ECG Results by Category and Visit (Safety Analysis Set) | 70 |
| Table 14.3-5.1 Physical Examination (Safety Analysis Set) | 71 |
| Table 14.3-6.1 NMP22 Test Results (Safety Analysis Set) | 72 |
| Listing 14.3-1.1 Deaths (Safety Analysis Set) | |
| Listing 14.3-2.1 Serious Non-fatal Adverse Events (Safety Analysis Set) | |
| Listing 14.3-3.1 Adverse Events Leading to Treatment Discontinuation (Safety Analysis Set) | 74 |
| Listing 14.3-4.1 Cardiovascular Adverse Events (Safety Analysis Set) | |
| Listing 14.3-5.1 Hypoglycemic Adverse Event (Safety Analysis Set) | 75 |
| Listing 14.3-6.1 Severe Hypoglycemic Adverse Events (Safety Analysis Set) | 76 |
| Listing 14.3-7.1 Renal and Urinary Adverse Events (Safety Analysis Set) | 76 |
| Listing 14.3-8.1 Genitourinary Adverse Events (Safety Analysis Set) | |
| Listing 14.3-9.1 Liver Adverse Events (Safety Analysis Set) | |
| Listing 14.3-10.1 Cancer Adverse Events (Safety Analysis Set) | |
| Listing 14.3-11.1 Bone Fracture Adverse Events (Safety Analysis Set) | |
| Listing 14.3-12.1 Clinically Significant Abnormal Hematology Laboratory Evaluations (Safety Analy | sis Set) 79 |
| Listing 14.3-12.2 Clinically Significant Abnormal Chemistry Laboratory Evaluations (Safety Analys | |
| Listing 14.3-12.3 Clinically Significant Abnormal Urinalysis Laboratory Evaluations (Safety Analy | |
| Listing 16.1-1.1 Randomized Allocation to Treatment (All Randomized Subjects) | |
| Listing 16.2-1.1 Subject Disposition (All Randomized Subjects) | |
| Listing 16.2-2.1 Inclusion/Exclusion Criteria Not Met (All Run-in Failures) | |
| Listing 16.2-2.2 Protocol Deviations (All Randomized Subjects) | |
| Listing 16.2-2.3 Major Protocol Deviations (All Randomized Subjects) | |
| Listing 16.2-3.1 Analysis Populations (All Randomized Subjects) | |
| Listing 16.2-4.1 Demographic Characteristics (Safety Analysis Set) | |
| Listing 16.2-4.2 Substance Use (Safety Analysis Set) | |
| Listing 16.2-4.3 Drug Screen Results (Safety Analysis Set) | |
| Listing 16.2-4.4 Medical History (Safety Analysis Set) | |
| Listing 16.2-4.5 Diabetes Medical History (Safety Analysis Set) | |
| Listing 16.2-5.1 Prior and Concomitant Medications (Safety Analysis Set) | 92 |

| Protocol: THR-1442-C-418 | Page x of y |
|---|---|
| Listing 16.2-6.1 Study Drug Administration (Safety Analysis Set) | 93 |
| Listing 16.2-7.1 HbA1c (%) (Full Analysis Set) | 94 |
| Listing 16.2-7.2 Fasting Plasma Glucose (mmol/L) (Full Analysis Set) | 95 |
| Listing 16.2-7.3 Weight(kg) (Full Analysis Set) | 95 |
| Listing 16.2-7.4 Systolic Blood Pressure (mmHg) (Full Analysis Set) | 96 |
| Listing 16.2-7.5 Diastolic Blood Pressure (mmHg) (Full Analysis Set) | 97 |
| Listing 16.2-8.1 Adverse Events (Safety Analysis Set) | 97 |
| Listing 16.2-8.2 Hypoglycemic Events Supplemental Information (Safety Analysis Set) | 98 |
| Listing 16.2-9.1 Hematology Laboratory Evaluations (Safety Analysis Set) | 99 |
| Listing 16.2-9.2 Chemistry Laboratory Evaluations (Safety Analysis Set) | 100 |
| Listing 16.2-9.3 Urinalysis Laboratory Evaluations (Safety Analysis Set) | 100 |
| Listing 16.2-10.1 Vital Signs (Safety Analysis Set) | |
| Listing 16.2-10.2 ECG Values (Safety Analysis Set) | 102 |
| Listing 16.2-10.3 Overall ECG Interpretations and Abnormal Findings (Safety Analysis Set) | 103 |
| Listing 16.2-10.4 Physical Examinations (Safety Analysis Set) | 104 |
| Listing 16.2-10.5 Pregnancies (Safety Analysis Set) | 105 |
| Listing 16.2-10.6 NMP22 Testing Results (Safety Analysis Set) | 106 |
Protocol: THR-1442-C-418 Page x of y

# Table 14.1-1.1.1 Subject Disposition for Run-in Failures (All Enrolled Subjects)

| | Total<br>(N=xxx) |
|-------------------------------------------------------|------------------|
| All Enrolled Subjects | xxx |
| All Randomized Subjects | xxx (xx.x%) |
| Discontinued Prior to Randomization (Run-in Failures) | xxx (xx.x%) |
| Reasons Discontinued Prior to Randomization | xxx (xx.x%) |
| Withdrew Consent | xxx (xx.x%) |
| Failed Inclusion/Exclusion Criteria | xxx (xx.x%) |
| Other | xxx (xx.x%) |
| XXXXXXXXXXXXXXXX | xxx (xx.x%) |

Note: Percentages are calculated using the number of subjects enrolled as the denominator.

Source Data: Listing 16.2-2.1

Table 14.1-1.1.2

Subject Disposition for Randomized Subjects

(All Randomized Subjects)

| | EGT0001442 | Placebo | Total |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Safety Analysis Set | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Full Analysis Set | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Per Protocol Analysis Set | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Completed Active Treatment through Week 24 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Discontuned Study before Week 24 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Reason for Discontinuing Study before Week 24 | | | |
| Clinically Significant Change in a Laboratory | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Investigator Terminates the Study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Patient Request to be Discontinued from the Study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Protocol Violation | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Serious or Intolerable Adverse Event | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Sponsor Termiantes the Study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXXXXXXXXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXXXXXXXXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Note: Percentages are calculated using the number of subjects randomized as the denominator.

Source Data: Listing 16.2-1.1

Table 14.1-1.1.2

Subject Disposition for Randomized Subjects

(All Randomized Subjects)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Completed Study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Discontinued Study Early | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Reason for Discontinuing Study Early | | | |
| Clinically Significant Change in a Laboratory | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Investigator Terminates the Study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Patient Request to be Discontinued from the Study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Protocol Violation | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Serious or Intolerable Adverse Event | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Sponsor Termiantes the Study | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXXXXXXXXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXXXXXXXXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Note: Percentages are calculated using the number of subjects randomized as the denominator.

Source Data: Listing 16.2-1.1

Protocol: THR-1442-C-418 Page x of y

# Table 14.1-1.1.3 Subject Disposition for Randomized Subjects by Country (All Randomized Subjects)

Same layout as Table 14.1-1.1.2. Display 'Country: United States' on the header of the table. Use the following footnote.

Note: Percentages are calculated using the number of subjects randomized as the denominator.

Source Data: Listing 16.2-1.1

Protocol: THR-1442-C-418 Page x of y

Table 14.1-1.2 Subjects Randomized by Country and Study Site (All Randomized Subjects)

| Country<br>Site | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| XXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Source Data: Listing 16.2-1.1

Protocol: THR-1442-C-418 Page x of y

## Table 14.1-1.3 Inclusion/Exclusion Criteria Not Met (All Run-in Failures)

Protocol Version Dated 2011-04-11

IN01:

IN02:

IN03:

···

EX01: EX02:

Protocol Versions Dated 2011-08-18, and 2011-09-12

IN01:

Note: All inclusion and exclusion criteria codes and full text are listed on page 1 of this summary.

Source Data: Listing 16.2-2.1

Protocol: THR-1442-C-418 Page x of y

## Table 14.1-1.3 Inclusion/Exclusion Criteria Not Met (All Run-in Failures)

| | Total<br>(N=xxx) |
|---|---|
| Subjects with Any Inclusion or Exclusion Criterion<br>Deviations | xxx (xx.x%) |
| Protocol Version Dated 2011-04-11<br>IN01 | xxx (xx.x%) |
| IN10 | xxx (xx.x%) |
| EX01 | xxx (xx.x%) |
| EX16 | xxx (xx.x%) |
| Protocol Versions Dated 2011-08-18, and 2011-09-12<br>IN01 | xxx (xx.x%) |
| IN10 | xxx (xx.x%) |
| EX01 | xxx (xx.x%) |
| EX19 | xxx (xx.x%) |

Note: All inclusion and exclusion criteria codes and full text are listed on page 1 of this summary. Source Data: Listing 16.2-2.1

Table 14.1-1.4.1
Demographics and Baseline Characteristics
(Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) | Total<br>(N=xxx) | p-value [1 |
|---|---|---|---|---|
| Age (years) | | | | 0.xxxx |
| n | xxx | xxx | XXX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | xx.x | xx.x | xx.x | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| Gender | | | | 0.xxxx |
| n | xxx | xxx | xxx | |
| Female | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Male | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Ethnicity | | | | 0.xxxx |
| n | xxx | xxx | xxx | |
| Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Not Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Child Bearing Potential | | | | 0.xxxx |
| n | xxx | xxx | xxx | |
| Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

<sup>[1]</sup> P-value is for testing the null hypotheses that summary statistics (mean or proportion) are equal among treatment groups. All tests are two-sided. \* indicates statistical significance at 0.05 level. Source Data: Listing 16.2-4.1

Table 14.1-1.4.1
Demographics and Baseline Characteristics
(Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) | Total<br>(N=xxx) | p-value [1] |
|---|---|---|---|---|
| Race | | | | 0.xxxx |
| n | xxx | xxx | xxx | |
| White or Caucasian | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Black or African American | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| American Indian or Alaskan Native | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Asian | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Native Hawaiian or Other Pacific Islander | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Baseline HbA1c Category | | | | 0.xxxx |
| n | xxx | xxx | xxx | |
| >=7% to <8.5% | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| >=8.5% to <=10% | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

<sup>[1]</sup> P-value is for testing the null hypotheses that summary statistics (mean or proportion) are equal among treatment groups. All tests are two-sided. \* indicates statistical significance at 0.05 level.

Source Data: Listing 16.2-4.1

Table 14.1-1.4.1

Demographics and Baseline Characteristics
(Safety Analysis Set)

| | EGT0001442 | Placebo | Total | |
|---|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) | p-value [1] |
| Height (cm) | | | | 0.xxxx |
| n | xxx | xxx | xxx | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | xx.x | xx.x | XX.X | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| Weight (kg) | | | | 0.xxxx |
| n | xxx | xxx | XXX | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | xx.x | xx.x | xx.x | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| Body Mass Index (BMI) (kg/m²) | | | | 0.xxxx |
| n | xxx | xxx | xxx | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| Median | xx.x | xx.x | XX.X | |
| Min, Max | xx, xx | xx, xx | xx, xx | |

<sup>[1]</sup> P-value is for testing the null hypotheses that summary statistics (mean or proportion) are equal among treatment groups. All tests are two-sided. \* indicates statistical significance at 0.05 level.

Source Data: Listing 16.2-4.1

Protocol: THR-1442-C-418 Page x of y

## Table 14.1-1.4.2 Demographics and Baseline Characteristics (Full Analysis Set)

Same layout as Table 14.1-1.4.1. Use the following footnote.

[1] P-value is for testing the null hypotheses that summary statistics (mean or proportion) are equal among treatment groups. All tests are two-sided. \* indicates statistical significance at 0.05 level.

Source Data: Listing 16.2-4.1

Table 14.1-1.4.3

Demographics and Baseline Characteristics
(Per Protocol Analysis Set)

Same layout as Table 14.1-1.4.1. Use the following footnote.

[1] P-value is for testing the null hypotheses that summary statistics (mean or proportion) are equal among treatment groups. All tests are two-sided. \* indicates statistical significance at 0.05 level.

Source Data: Listing 16.2-4.1

Table 14.1-1.4.4

Demographics and Baseline Characteristics by Country
(Safety Analysis Set)

Same layout as Table 14.1-1.4.1. Display 'Country: United States' on the header of the table. Use the following footnote.

[1] P-value is for testing the null hypotheses that summary statistics (mean or proportion) are equal among treatment groups. All tests are two-sided. \* indicates statistical significance at 0.05 level.

Source Data: Listing 16.2-4.1

Table 14.1-1.5 Substance Use (Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) | Total (N=xxx) |
|---|---|---|---|
| Alcohol Consumption | xxx | xxx | xxx |
| n | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | | | |
| Alcohol Units Consumed Per Week | | | |
| n | xxx | xxx | xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Tobacco Use | | | |
| n | xxx | XXX | XXX |
| Never Used | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Current User | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Former User | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Drug Dependency or Abuse | xxx | xxx | xxx |
| n | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | | | |

Source Data: Listing 16.2-4.2

Protocol: THR-1442-C-418 Page x of y

Table 14.1-2.1 Medical History (Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|------------------------------|-----------------------|--------------------|
| Subjects with Any Conditions | xxx (xx.x%) | xxx (xx.x%) |
| xxxxxxx | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXXX | xxx (xx.x%) | xxx (xx.x%) |
| OTHER | xxx (xx.x%) | xxx (xx.x%) |

Source Data: Listing 16.2-4.4

### Table 14.1-2.2 Diabetes Disease History (Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|---|---|---|
| Duration of Diabetes (years) [1] | | |
| n | xxx | xxx |
| Mean (SD) | xx.x (xx.xxx) | xx.x (xx.xxx) |
| Median | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx |
| Baseline Diabetes Therapy | | |
| n | xxx | XXX |
| Treatment Naive | xxx (xx.x%) | xxx (xx.x%) |
| Treated with One Anti-diabetic Agent | xxx (xx.x%) | xxx (xx.x%) |
| Blindness | | |
| n | xxx | xxx |
| Yes | xxx (xx.x%) | xxx (xx.x%) |
| No | xxx (xx.x%) | xxx (xx.x%) |
| Cataracts | | |
| Retinopathy | | |
| Laser Treatment to Either Eye | | |
| Foot Ulceration | | |
| Peripheral Neuropathy | | |
| Lower Limb Amputation | | |
| Diabetic Nephropathy | | |
| Current Microalbuminuria | | |
| Current Proteinuria | | |
| Dialysis | | |
| Kidney Transplantation | | |
| Major Hypoglycemic Event | | |
| Documented Hypoglycemic Event | | |

<sup>[1]</sup> To calculate duration from a partial diagnosis date, a missing month is imputed as January and a missing day is imputed as the first of the month.

Source Data: Listings 16.2-4.4 and 16.2-4.5

Protocol: THR-1442-C-418 Page x of y

## Table 14.1-2.3 Diabetes Disease History by Country (Safety Analysis Set)

Same layout as Table 14.1-2.3. Display 'Country: United States' on the header of the table. Use the following footnote

[1] To calculate duration from a partial diagnosis date, a missing month is imputed as January and a missing day is imputed as the first of the month.

Source Data: Listings 16.2-4.4 and 16.2-4.5

<DIRECTORY PATH>PROGRAM NAME Executed: DDMMMYYYY hh:mm Data Extracted: DDMONYYYY

Final - 22November2011 

Table 14.1-3.1 Prior Medications (Safety Analysis Set)

| TC Level 4 Term Preferred Term | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|--------------------------------|-----------------------|--------------------|
| Subjects with Any Medications | xxx (xx.x%) | xxx (xx.x%) |
| TC Level 4 Term #1 | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #1 | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #2 | xxx (xx.x%) | xxx (xx.x%) |
| TC Level 4 Term #2 | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) |

Note: At each level of summarization, a subject is counted once if the subject reported one or more medications.

Medications are coded using WHODRUG enhanced version June 2011. Prior medications are those started before the first dose of study medication.

Source Data: Listing 16.2-5.1

Table 14.1-3.2 Concomitant Medications (Safety Analysis Set)

| TC Level 4 Term<br>Preferred Term | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|---|---|---|
| ubjects with Any Medications | xxx (xx.x%) | xxx (xx.x%) |
| TC Level 4 Term #1 | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #1 | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #2 | xxx (xx.x%) | xxx (xx.x%) |
| TC Level 4 Term #2 | xxx (xx.x%) | xxx (xx.x%) |
| XXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXX | xxx (xx.x%) | xxx (xx.x%) |

Note: At each level of summarization, a subject is counted once if the subject reported one or more medications.

Medications are coded using WHODRUG enhanced version June 2011. Concomitant medications are those taken at any time on or after the day of the first dose of study medication, including those started prior to randomization but were continuing during the study period.

Source Data: Listing 16.2-5.1

Protocol: THR-1442-C-418 Page x of y

Table 14.1-3.3
Hyperglycemia Rescue Medications
(Safety Analysis Set)

| ATC Level 4 Term Preferred Term | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|---|---|---|
| rielelied leim | (IV-XXX) | (N-XXX) |
| Subjects with Any Rescue Medications | xxx (xx.x%) | xxx (xx.x%) |
| ATC Level 4 Term #1 | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #1 | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #2 | xxx (xx.x%) | xxx (xx.x%) |
| ATC Level 4 Term #2 | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) |
| XXXXXX | xxx (xx.x%) | xxx (xx.x%) |

Note: Only concomitant anti-hyperglycemia medications that are indicated by the investigator as being used for hyperglycemia rescue are included in this summary. At each level of summarization, a subject is counted once if the subject reported one or more medications. Medications are coded using WHODRUG enhanced version June 2011. Concomitant rescue medications are those taken at any time on or after the day of the first dose of study medication.

Source Data: Listing 16.2-5.1

Table 14.1-3.4

Proportion of Subjects with Hyperglycemia Rescue (Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|---|---|---|
| umber of Subjects Rescued by Time of First Rescue | | |
| <=2 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >2 weeks - <=6 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >6 weeks - <=12 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >12 weeks - <=18 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >18 weeks - <=24 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >24 weeks - <=36 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >36 weeks - <=48 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >48 weeks - <=60 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >60 weeks - <=72 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >72 weeks - <=84 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >84 weeks - <=96 weeks | xxx (xx.x%) | xxx (xx.x%) |

Source Data: Listing 16.2-5.1

Table 14.1-4.1 Treatment Exposure (Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo |
|---|---|---|
| | | (N=xxx) |
| Ouration of Exposure (weeks) | | |
| n | xxx | xxx |
| Mean (SD) | xx.x (xx.xxx) | xx.x (xx.xxx) |
| Median | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx |
| Jumber (%) of Subjects with Exposure of | | |
| 1 Dose | xxx (xx.x%) | xxx (xx.x%) |
| >1 Dose - <=2 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >2 weeks - <=6 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >6 weeks - <=12 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >12 weeks - <=18 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >18 weeks - <=24 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >24 weeks - <=36 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >36 weeks - <=48 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >48 weeks - <=60 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >60 weeks - <=72 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >72 weeks - <=84 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >84 weeks - <=96 weeks | xxx (xx.x%) | xxx (xx.x%) |
| >96 weeks | xxx (xx.x%) | xxx (xx.x%) |

Note: Duration of exposure (weeks) =  $(date\ of\ last\ dose\ -\ date\ of\ first\ dose\ +\ 1)/7.$ 

Source Data: Listing 16.2-6.1

Protocol: THR-1442-C-418 Page x of y

Table 14.1-4.2 Treatment Compliance (Safety Analysis Set)

| | EGT0001442 | Placebo |
|---------------------|---------------|---------------|
| | (N=xxx) | (N=xxx) |
| Compliance (%) | | |
| n | XXX | xxx |
| Mean (SD) | xx.x (xx.xxx) | xx.x (xx.xxx) |
| Median | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx |
| Compliance Category | | |
| n | XXX | xxx |
| <80% | xxx (xx.x%) | xxx (xx.x%) |
| >=80% | xxx (xx.x%) | xxx (xx.x%) |

Note: Treatment compliance is calculated as total number of administered capsules divided by total number of capsules which should have been taken based on the last completed visit during active treatment period.

Source Data: Listing 16.2-6.1





Source Data: Table 14.2-1.3

Programming Note: Display treatment group identifiers identical to those in summary tables instead of using TRT A and TRT B as shown in the shell. Also, this shell only shows through Week 52 but our data and plot will go through Week 97.

Protocol: THR-1442-C-418 Page x of y

Figure 14.2-1.2
Line Graph of Mean (+/- SE) HbAlc (%), Excluding Post-Rescue Values
(Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-1.3

Figure 14.2-2.1

Line Graph of Mean (+/-SE) Change from Baseline in Fasting Plasma Glucose (mmol/L), Excluding Post-Rescue Values (Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-2.3

Figure 14.2-2.2

Line Graph of Mean (+/- SE) Fasting Plasma Glucose (mmol/L), Excluding Post-Rescue Values (Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-2.3

Protocol: THR-1442-C-418 Page x of y

Figure 14.2-3.1

Line Graph of Mean (+/- SE) Change from Baseline in Weight (kg), Excluding Post-Rescue Values (Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-3.3

Figure 14.2-3.2

Line Graph of Mean (+/- SE) Weight (kg), Excluding Post-Rescue Values (Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-3.3

Figure 14.2-4.1

Line Graph of Mean (+/- SE) Change from Baseline in Systolic Blood Pressure (mmHg), Excluding Post-Rescue Values (Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-4.3

Protocol: THR-1442-C-418 Page x of y

Figure 14.2-4.2

Line Graph of Mean (+/- SE) Systolic Blood Pressure (mmHg), Excluding Post-Rescue Values (Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-4.3

Figure 14.2-5.1

Line Graph of Mean (+/- SE) Change from Baseline in Diastolic Blood Pressure (mmHg), Excluding Post-Rescue Values (Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-5.3

Figure 14.2-5.2

Line Graph of Mean (+/- SE) Diastolic Blood Pressure (mmHg), Excluding Post-Rescue Values (Full Analysis Set - OC)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.2-5.3

## Table 14.2-1.1 Analysis of Change from Baseline in HbA1c (%) at Week 24 (Full Analysis Set - LOCF)

Week 24

| | EGT0001442 | Placebo |
|-----------------------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| Number of Subjects [1] | xxx | xxx |
| Number (%) of Values Carried Forward | xx (xx.x%) | xx (xx.x%) |
| Baseline | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Week 24 | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| p-value [2] | 0.xxxx | |
| Model-Adjusted Change from Baseline [3] | | |
| LS Mean (SE) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| 95% Confidence Interval | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Difference from Placebo [3] | | |
| Difference of LS Means | xx.xx | |
| 95% Confidence Interval | (xx.xx, xx.xx) | |
| p-value | 0.xxxx | |

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline HbAlc + site + age category + gender + race.

Source Data: Listing 16.2-7.1

Table 14.2-1.2

Analysis of Change from Baseline in HbA1c (%)
(Full Analysis Set - LOCF)

Week 2

| | EGT0001442 | Placebo |
|-----------------------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| Number of Subjects [1] | xxx | xxx |
| Number (%) of Values Carried Forward | xx (xx.x%) | xx (xx.x%) |
| Baseline | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Week 2 | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| p-value [2] | 0.xxxx | |
| Model-Adjusted Change from Baseline [3] | | |
| LS Mean (SE) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| 95% Confidence Interval | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Difference from Placebo [3] | | |
| Difference of LS Means | xx.xx | |
| 95% Confidence Interval | (xx.xx, xx.xx) | |
| p-value | 0.xxxx | |

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline HbAlc + site + age category + gender + race.

Source Data: Listing 16.2-7.1

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Table 14.2-1.3

Analysis of Change from Baseline in HbA1c (%), Excluding Post-Rescue Values (Full Analysis Set - OC)

Week 2

| | EGT0001442 | Placebo |
|-----------------------------------------|----------------|----------------|
| | (N=xxx) | (N=xxx) |
| Number of Subjects [1] | xxx | xxx |
| Baseline | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Week 2 | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| p-value [2] | 0.xxxx | |
| Model-Adjusted Change from Baseline [3] | | |
| LS Mean (SE) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| 95% Confidence Interval | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Difference from Placebo [3] | | |
| Difference of LS Means | xx.xx | |
| 95% Confidence Interval | (xx.xx, xx.xx) | |
| p-value | 0.xxxx | |

Note: This analysis uses observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline HbAlc + site + age category + gender + race.

Source Data: Listing 16.2-7.1

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Table 14.2-1.4

Repeated Measures Analysis of Change from Baseline in HbAlc (%) at Week 96, Excluding Post-rescue Values (Full Analysis Set - OC)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|---|---|---|
| Model-Adjusted Change from Baseline at Week 96 [1] | | |
| n (# of Subjects) | xx | xx |
| k (# of Post-baseline Visits) | xx | xx |
| LS Mean (SE) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| 95% Confidence Interval | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Difference from Placebo [1] | | |
| Difference of LS Means | xx.xx | |
| 95% Confidence Interval | (xx.xx, xx.xx) | |
| p-value | 0.xxxx | |

Note: This analysis uses all observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

Source Data: Listing 16.2-7.1

 $<sup>\</sup>ensuremath{\texttt{[1]}}$  Based on repeated measure model including treatment and visit as factors.

Protocol: THR-1442-C-418 Page x of y

## Table 14.2-1.5 Summary Statistics for HbA1c (%) (Full Analysis Set - OC)

Screening

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|------------------------|-----------------------|--------------------|
| Number of Subjects [1] | xxx | xxx |
| Screening<br>Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | XX.XX | XX.XX |
| Min, Max | xx.x, xx.x | xx.x, xx.x |

Note: This summary uses all observed values; no missing data imputation is performed. Baseline is defined as the last available assessment on or prior to the first dose of study drug.

[1] For Screening and Week 0 the number of subjects with a value at the specified visit is displayed. For all post-baseline visits, the number of subjects with a value at baseline and at the specified visit is displayed. Source Data: Listing 16.2-7.1

Programming Note: Use page 1 shell for Screening and Week 0, use pages 2 shell for the remaining post-baseline visits (Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up).

Protocol: THR-1442-C-418 Page x of y

Table 14.2-1.5

Summary Statistics for HbA1c (%)

(Full Analysis Set - OC)

Week 2

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|------------------------|-----------------------|--------------------|
| Number of Subjects [1] | xxx | xxx |
| Baseline | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Week 2 | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | xx.xx | xx.xx |
| Min, Max | XX.X, XX.X | xx.x, xx.x |

Note: This summary uses all observed values; no missing data imputation is performed. Baseline is defined as the last available assessment on or prior to the first dose of study drug.

[1] For Screening and Week 0 the number of subjects with a value at the specified visit is displayed. For all post-baseline visits, the number of subjects with a value at baseline and at the specified visit is displayed. Source Data: Listing 16.2-7.1

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

### Table 14.2-1.6 Analysis of Change from Baseline in HbA1c (%) (Per Protocol Analysis Set - LOCF)

Programming Note: See Table 14.2-1.1 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline HbAlc + site + age category + gender + race.

Source Data: Listing 16.2-7.1

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Table 14.2-2.1 Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L) at Week 24 (Full Analysis Set - LOCF)

Programming Note: See Table 14.2-1.1 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline FPG + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.2

Protocol: THR-1442-C-418 Page x of y

#### Table 14.2-2.2

Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L) (Full Analysis Set - LOCF)

Programming Note: See Table 14.2-1.2 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline FPG + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.2

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

#### Table 14.2-2.3

Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L), Excluding Post-rescue Values (Full Analysis Set- OC)

#### Programming Note: See Table 14.2-1.3 for layout. Use footnotes below.

Note: This analysis uses observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline FPG + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.2

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

#### Table 14.2-2.4

Repeated Measures Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L) at Week 96, Excluding Post-rescue Values

(Full Analysis Set - OC)

Programming Note: See Table 14.2-1.4 for layout. Use footnotes below.

Note: This analysis uses all observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

[1] Based on repeated measure model including treatment and visit as factors.

Source Data: Listing 16.2-7.2

Protocol: THR-1442-C-418 Page x of y

#### Table 14.2-2.5 Summary Statistics for Fasting Plasma Glucose (mmol/L) (Full Analysis Set- OC)

Programming Note: See Table 14.2-1.5 for layout. Use footnotes below.

Note: This summary uses all observed values; no missing data imputation is performed. Baseline is defined as the last available assessment on or prior to the first dose of study drug.

[1] For Screening and Week 0 the number of subjects with a value at the specified visit is displayed. For all post-baseline visits, the number of subjects with a value at baseline and at the specified visit is displayed. Source Data: Listing 16.2-7.2

Programming Note: Use page 1 shell for Screening and Week 0, use pages 2 shell for the remaining post-baseline visits (Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up).

### Table 14.2-2.6 Analysis of Change from Baseline in Fasting Plasma Glucose (mmol/L) (Per Protocol Analysis Set - LOCF)

Programming Note: See Table 14.2-1.2 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline FPG + baseline HbA1c category + site + age category + gender + race. Source Data: Listing 16.2-7.2

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

### Table 14.2-3.1 Analysis of Change from Baseline in Weight (kg) at Week 24 (Full Analysis Set - LOCF)

Programming Note: See Table 14.2-1.1 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline weight + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.3

Table 14.2-3.2

Analysis of Change from Baseline in Weight (kg)

(Full Analysis Set - LOCF)

Programming Note: See Table 14.2-1.2 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline weight + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.3

Programming Note: present for Weeks 12, 24, 48, 72, 96, 97 and 1 week follow-up.
Protocol: THR-1442-C-418 Page x of y

#### Table 14.2-3.3

Analysis of Change from Baseline in Weight (kg), Excluding Post-rescue Values (Full Analysis Set- OC)

Programming Note: See Table 14.2-1.3 for layout. Use footnotes below.

Note: This analysis uses observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline weight + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.3

Programming Note: present for Weeks 12, 24, 48, 72, 96, 97 and 1 week follow-up.

### Table 14.2-3.4

Repeated Measures Analysis of Change from Baseline in Weight (kg) at Week 96, Excluding Post-rescue Values (Full Analysis Set - OC)

Programming Note: See Table 14.2-1.4 for layout. Use footnotes below.

Note: This analysis uses all observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

[1] Based on repeated measure model including treatment and visit as factors.

Source Data: Listing 16.2-7.3

Protocol: THR-1442-C-418 Page x of y

## Table 14.2-3.5 Summary Statistics for Weight (kg) (Full Analysis Set- OC)

Programming Note: See Table 14.2-1.5 for layout. Use footnotes below.

Note: This summary uses all observed values; no missing data imputation is performed. Baseline is defined as the last available assessment on or prior to the first dose of study drug.

[1] For Screening and Week 0 the number of subjects with a value at the specified visit is displayed. For all post-baseline visits, the number of subjects with a value at baseline and at the specified visit is displayed. Source Data: Listing 16.2-7.3

Programming Note: use page 1 shell for Screening, and use page 2 shell for the remaining post-baseline visits (Weeks 12, 24, 48, 72, 96, 97 and 1 week follow-up).

# Table 14.2-3.6 Analysis of Change from Baseline in Weight (kg) (Per Protocol Analysis Set - LOCF)

Programming Note: See Table 14.2-1.2 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline weight + baseline HbA1c category + site + age category + gender + race. Source Data: Listing 16.2-7.3

Programming Note: present for Weeks 12, 24, 48, 72, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

### Table 14.2-4.1

Analysis of Change from Baseline in Systolic Blood Pressure (mmHg) at Week 24 (Full Analysis Set - LOCF)

Programming Note: See Table 14.2-1.1 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline SBP + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.4

Table 14.2-4.2

Analysis of Change from Baseline in Systolic Blood Pressure (mmHg)

(Full Analysis Set - LOCF)

Programming Note: See Table 14.2-1.2 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline SBP + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.4

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

Table 14.2-4.3

Analysis of Change from Baseline in Systolic Blood Pressure (mmHg), Excluding Post-rescue Values (Full Analysis Set- OC)

Programming Note: See Table 14.2-1.3 for layout. Use footnotes below.

Note: This analysis uses observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline SBP + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.4

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Table 14.2-4.4

Repeated Measures Analysis of Change from Baseline in Systolic Blood Pressure (mmHg) at Week 96, Excluding Post-rescue Values

(Full Analysis Set - OC)

Programming Note: See Table 14.2-1.4 for layout. Use footnotes below.

Note: This analysis uses all observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

[1] Based on repeated measure model including treatment and visit as factors.

Source Data: Listing 16.2-7.4

Protocol: THR-1442-C-418 Page x of y

# Table 14.2-4.5 Summary Statistics for Systolic Blood Pressure (mmHg) (Full Analysis Set- OC)

Programming Note: See Table 14.2-1.5 for layout. Use footnotes below.

Note: This summary uses all observed values; no missing data imputation is performed. Baseline is defined as the last available assessment on or prior to the first dose of study drug.

[1] For Screening and Week 0 the number of subjects with a value at the specified visit is displayed. For all post-baseline visits, the number of subjects with a value at baseline and at the specified visit is displayed. Source Data: Listing 16.2-7.4

Programming Note: Use page 1 shell for Screening, Week -2 and Week 0, use pages 2 shell for the remaining post-baseline visits (Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up).

# Table 14.2-4.6 Analysis of Change from Baseline in Systolic Blood Pressure (mmHg) (Per Protocol Analysis Set - LOCF)

Programming Note: See Table 14.2-1.2 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline SBP + baseline HbA1c category + site + age category + gender + race. Source Data: Listing 16.2-7.4

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

### Table 14.2-5.1

Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg) at Week 24 (Full Analysis Set - LOCF)

Programming Note: See Table 14.2-1.1 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline DBP + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.5

# Table 14.2-5.2 Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg) (Full Analysis Set - LOCF)

Programming Note: See Table 14.2-1.2 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline DBP + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.5

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

### Table 14.2-5.3

Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg), Excluding Post-rescue Values (Full Analysis Set- OC)

Programming Note: See Table 14.2-1.3 for layout. Use footnotes below.

Note: This analysis uses observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline DBP + baseline HbA1c category + site + age category + gender + race.

Source Data: Listing 16.2-7.5

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

### Table 14.2-5.4

Repeated Measures Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg) at Week 96, Excluding Post-rescue Values

(Full Analysis Set - OC)

Programming Note: See Table 14.2-1.4 for layout. Use footnotes below.

Note: This analysis uses all observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

[1] Based on repeated measure model including treatment and visit as factors.

Source Data: Listing 16.2-7.5

Protocol: THR-1442-C-418 Page x of y

## Table 14.2-5.5 Summary Statistics for Diastolic Blood Pressure (mmHg) (Full Analysis Set- OC)

Programming Note: See Table 14.2-1.5 for layout. Use footnotes below.

Note: This summary uses all observed values; no missing data imputation is performed. Baseline is defined as the last available assessment on or prior to the first dose of study drug.

[1] For Screening and Week 0 the number of subjects with a value at the specified visit is displayed. For all post-baseline visits, the number of subjects with a value at baseline and at the specified visit is displayed. Source Data: Listing 16.2-7.5

Programming Note: Use page 1 shell for Screening, Week -2 and Week 0, use pages 2 shell for the remaining post-baseline visits (Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up).

## Table 14.2-5.6 Analysis of Change from Baseline in Diastolic Blood Pressure (mmHg) (Per Protocol Analysis Set - LOCF)

Programming Note: See Table 14.2-1.2 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a two-sided t-test for the difference in means of change from baseline.
- [3] Based on ANCOVA: Change = trt + baseline DBP + baseline HbA1c category + site + age category + gender + race. Source Data: Listing 16.2-7.5

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Table 14.2-6.1
Analysis of Proportion of Subjects Achieving HbAlc <7%
(Full Analysis Set- LOCF)

| | EGT0001442 | Placebo |
|--------------------------------------|------------|------------|
| | (N=xxx) | (N=xxx) |
| eek 2 | | |
| Number of Subjects [1] | xxx | xxx |
| Number (%) of Values Carried Forward | xx (xx.x%) | xx (xx.x%) |
| Subjects Achieving HbA1c <7% | xx (xx.x%) | xx (xx.x%) |
| p-value [2] | 0.xxxx | |
| eek 6 | | |
| Number of Subjects [1] | xxx | xxx |
| Number (%) of Values Carried Forward | xx (xx.x%) | xx (xx.x%) |
| Subjects Achieving HbA1c <7% | xx (xx.x%) | xx (xx.x%) |
| p-value [2] | 0.xxxx | |
| eek 12 | | |
| Number of Subjects [1] | xxx | xxx |
| Number (%) of Values Carried Forward | xx (xx.x%) | xx (xx.x%) |
| Subjects Achieving HbA1c <7% | xx (xx.x%) | xx (xx.x%) |
| p-value [2] | 0.xxxx | |

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a chi-square test for the difference in proportions.

Source Data: Listing 16.2-7.1

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Table 14.2-6.2
Analysis of Proportion of Subjects Achieving HbAlc <7%, Excluding Post-Rescue Values (Full Analysis Set- OC)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|------------------------------|-----------------------|--------------------|
| eek 2 | | |
| Number of Subjects [1] | xxx | xxx |
| Subjects Achieving HbA1c <7% | xx (xx.x%) | xx (xx.x%) |
| p-value [2] | 0.xxxx | |
| eek 6 | | |
| Number of Subjects [1] | xxx | xxx |
| Subjects Achieving HbA1c <7% | xx (xx.x%) | xx (xx.x%) |
| p-value [2] | 0.xxxx | |
| ek 12 | | |
| Number of Subjects [1] | xxx | xxx |
| Subjects Achieving HbA1c <7% | xx (xx.x%) | xx (xx.x%) |
| p-value [2] | 0.xxxx | |

Note: This analysis uses observed values excluding those obtained after hyperglycemia rescue; no missing data imputation is performed. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a chi-square test for the difference in proportions.

Source Data: Listing 16.2-7.1

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

Table 14.2-6.3

Summary Statistics for Proportion of Subjects Achieving HbAlc <7% by Visit

(Full Analysis Set- OC)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|-----------|-----------------------|--------------------|
| Gcreening | xxx (xx.x%) | xxx (xx.x%) |
| Jeek 0 | xxx (xx.x%) | xxx (xx.x%) |
| Jeek 2 | xxx (xx.x%) | xxx (xx.x%) |
| Jeek 6 | xxx (xx.x%) | xxx (xx.x%) |
| Jeek 12 | xxx (xx.x%) | xxx (xx.x%) |

Note: This analysis uses all observed values; no missing data imputation is performed. Source Data: Listing 16.2-7.1

Programming Note: present for Screening, Weeks 0, 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

# Table 14.2-6.4 Analysis of Proportion of Subjects Achieving HbA1c <7% (Per Protocol Analysis Set- LOCF)

Programming Note: See Table 14.2-6.1 for layout. Use footnotes below.

Note: This analysis uses the last observation carried forward (LOCF) method for missing post-baseline values as well as for values obtained after hyperglycemia rescue. \* indicates statistical significance at 0.05 level.

- [1] Number of subjects with a value at baseline and at the specified visit.
- [2] The p-value is from a chi-square test for the difference in proportions.

Source Data: Listing 16.2-7.1

Programming Note: present for Weeks 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

Figure 14.3-2.1
Line Graph of Mean (+/- SE) Results for Hematology (Safety Analysis Set)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.3-2.1

Figure 14.3-2.2
Line Graph of Mean (+/- SE) Results for Chemistry (Safety Analysis Set)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.3-2.2

Protocol: THR-1442-C-418 Page x of y

Figure 14.3-3.1
Line Graph of Mean (+/- SE) Results for Vital Signs (Safety Analysis Set)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.3-3.1

Figure 14.3-4.1
Line Graph of Mean (+/- SE) ECG Results
(Safety Analysis Set)

See Figure 14.2-1.1 for layout and general programming notes. Use footnotes below.

Source Data: Table 14.3-4.1

Table 14.3-1.1

Overall Summary of Adverse Events
(Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Number of Subjects with at Least One AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects With at Least One TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects With at Least One Treatment-<br>related TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects With at Least One Serious TEAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects With at Least One TEAE Leading to Treatment Discontinuation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects With at Least One TEAE Leading to Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: For each level of summarization, a subject is counted once if the subject reported one or more events. Percentages are based on the number of subjects in each treatment group.

Source Data: Listing 16.2-8.1

Table 14.3-1.2
Treatment Emergent Adverse Events
(Safety Analysis Set)

| System Organ Class Preferred Term | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Total Number of Events | xx | xx | xx |
| Number of Subjects With at Least One Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| System Organ Class #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: For each level of summarization, a subject is counted once if the subject reported one or more events.

Percentages are based on the number of subjects in each treatment group. The system organ class (SOC) and preferred term within the SOC are presented by decreasing frequency of incidence for all treatment groups combined.

Source Data: Listing 16.2-8.1

Protocol: THR-1442-C-418

Table 14.3-1.3

Treatment Emergent Adverse Events by Severity
(Safety Analysis Set)

Page x of y

| Preferred Term | EGT0001442 | Placebo | Total |
|---|---|---|---|
| Severity | (N=xxx) | (N=xxx) | (N=xxx) |
| Number of Subjects With at Least One Event | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| System Organ Class #1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #2 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Note: AEs with missing severity are considered severe in this summary. Percentages are based on the number of subjects in each treatment group. For each level of summarization, a subject is counted once according to the maximum severity experienced if the subject reported one or more events. The system organ class (SOC) and preferred term within the SOC are presented by decreasing frequency of incidence for all treatment groups combined.

Source Data: Listing 16.2-8.1

Programming Note: Only display severity level rows if there are subjects who have experienced that maximum severity level. Present SOC and PT within SOC by decreasing frequency of overall incidence. (Sort order should match 14.3-1.1)

Table 14.3-1.4

Treatment Emergent Adverse Events by Relationship to Study Drug (Safety Analysis Set)

| System Organ Class | | | |
|---|---|---|---|
| Preferred Term | EGT0001442 | Placebo | Total |
| Relationship to Study Drug | (N=xxx) | (N=xxx) | (N=xxx) |
| Number of Subjects With at Least One Event | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| System Organ Class #1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Preferred Term #2 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| • • • | | | |

Note: Related includes the relationship judged by investigators as possible, probable, and definite. Not related includes not related and unlikely. AEs with missing relationship to study drug are considered related in this summary. For each level of summarization, a subject is counted once according to the greatest relationship to study drug if the subject reported one or more events. Percentages are based on the number of subjects in each treatment group. The system organ class (SOC) and preferred term within the SOC are presented by decreasing frequency of incidence for all treatment groups combined.

Source Data: Listing 16.2-8.1

Programming Note: Only display relationship rows if there are subjects who have experienced that maximum intensity level. Present SOC and PT within SOC by decreasing frequency of overall incidence. (Sort order should match 14.3-1.1)

Protocol: THR-1442-C-418 Page x of y

# Table 14.3-1.5 Most Common Treatment Emergent Adverse Events (Safety Analysis Set)

### See Table 14.3-1.1 for layout. Use footnotes below.

Note: This summary presents AEs that occur in >5% of the subjects in either of the treatment groups. For each level of summarization, a subject is counted once if the subject reported one or more events. Percentages are based on the number of subjects in each treatment group. The system organ class (SOC) and preferred term within the SOC are presented by decreasing frequency of incidence for all treatment groups combined.

Source Data: Listing 16.2-8.1

Table 14.3-1.6
Serious Treatment Emergent Adverse Events
(Safety Analysis Set)

### See Table 14.3-1.1 for layout. Use footnotes below.

Note: For each level of summarization, a subject is counted once if the subject reported one or more events.

Percentages are based on the number of subjects in each treatment group. The system organ class (SOC) and preferred term within the SOC are presented by decreasing frequency of incidence for all treatment groups combined.

Source Data: Listing 16.2-8.1

Protocol: THR-1442-C-418 Page x of y

### Table 14.3-1.7

Treatment Emergent Adverse Events Leading to Treatment Discontinuation (Safety Analysis Set)

See Table 14.3-1.1 for layout. Use footnotes below.

Note: For each level of summarization, a subject is counted once if the subject reported one or more events.

Percentages are based on the number of subjects in each treatment group. The system organ class (SOC) and preferred term within the SOC are presented by decreasing frequency of incidence for all treatment groups combined.

Source Data: Listing 16.2-8.1

Table 14.3-1.8

Treatment Emergent Hypoglycemic Events by Severity and Intervention (Safety Analysis Set)

| | EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Total Number of Events | xx | xx | xx |
| Number of Subjects With at Least One Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severity | | | |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Documented Symptomatic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Asymptomatic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Probable Symptomatic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Relative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Intervention [1] | | | |
| Extensive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Immediate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Minor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Missing | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: For each level of summarization, a subject is counted in all severity or intervention categories if the subject reported one or more events. Percentages are based on the number of subjects in each treatment group.

Source Data: Listing 16.2-8.1

<sup>[1]</sup> Extensive = glucose injection/infusion/glucagon; Immediate = glucose drinks or supplements; Minor = administered sugary drinks or sweets; None = no intervention.

Table 14.3-2.1 Change from Baseline in Hematology (Safety Analysis Set)

| | EGT00 | 01442 | Plac | cebo |
|---|---|---|---|---|
| | (N=xxx) | | (N=2 | xxx) |
| | | Change from | | Change from |
| | Result | Baseline | Result | Baseline |
| Lab Test #1 (unit) | | | | |
| Baseline | | | | |
| n | xxx | | xxx | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | |
| Week 2 | | | | |
| n | xxx | xxx | xxx | xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |

Note: Baseline is defined as the last available assessment on or prior to the first dose of study medication. Source Data: Listing 16.2-9.1

Programming note: use timepoints of Baseline, Week 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

## Table 14.3-2.2 Change from Baseline in Chemistry (Safety Analysis Set)

See table 14.3-2.1 for layout. Use footnote below.

Note: Baseline is defined as the last available assessment on or prior to the first dose of study medication. Source Data: Listing 16.2-9.2

Programming note: use timepoints of Baseline, Week 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

<DIRECTORY PATH>PROGRAM NAME Executed: DDMMMYYYY hh:mm Data Extracted: DDMONYYYY

Final - 22November2011 

Table 14.3-2.3 Urinalysis (Safety Analysis Set)

| | EGT0001442 | Placebo |
|-----------------|--------------|--------------|
| | (N=xxx) | (N=xxx) |
| Albumin (unit) | | |
| Screening | | |
| n | xxx | xxx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx |
| Week 0 | | |
| Urinary Protein | | |
| Screening | | |
| n | xxx (xx.x%) | xxx (xx.x%) |
| 4 | xxx (xx.x%) | xxx (xx.x%) |
| 5 | xxx (xx.x%) | xxx (xx.x%) |
| · | | |

Source Data: Listing 16.2-9.3

Programming note: use timepoints of Screening, Week 0, 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

Table 14.3-2.4 Shift in Hematology (Safety Analysis Set)

| | | EGT0001442 | | | Placebo | |
|---|---|---|---|---|---|---|
| | (N=xxx) | | (N=xxx) | | | |
| | | Baseline | | | Baseline | |
| | Low | Normal | High | Low | Normal | High |
| Lab Test #1 (unit) | | | | | | |
| Week 2 | | n = xxx | | | n = xxx | |
| Low | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Normal | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| High | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Week 6 | | n = xxx | | | n = xxx | |
| Low | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Normal | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| High | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Note: Baseline is defined as the last available assessment on or prior to the first dose of study medication. The number of subjects with a value at baseline and at the specified visit is displayed.

Source Data: Listing 16.2-9.1

Programming note: use all available timepoints per data following order such as Baseline, Week 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

Table 14.3-2.5 Shift in Chemistry (Safety Analysis Set)

### See table 14.3-2.4 for layout. Use footnotes below.

Note: Baseline is defined as the last available assessment on or prior to the first dose of study medication. The number of subjects with a value at baseline and at the specified visit is displayed.

Source Data: Listing 16.2-9.2

Programming note: use all available timepoints per data following order such as Baseline, Week 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Table 14.3-2.6 Shift in Urinalysis (Safety Analysis Set)

### See table 14.3-2.4 for layout. Use footnotes below.

Note: Baseline is defined as the last available assessment on or prior to the first dose of study medication. The number of subjects with a value at baseline and at the specified visit is displayed.

Source Data: Listing 16.2-9.3

Programming note: use all available timepoints per data following order such as Baseline, Week 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up.

Protocol: THR-1442-C-418 Page x of y

Table 14.3-3.1 Change from Baseline in Vital Signs (Safety Analysis Set)

See table 14.3-2.1 for layout. Use footnote below.

Note: Baseline is defined as the last available assessment on or prior to the first dose of study medication. Source Data: Listing 16.2-10.1

Programming note: use timepoints of Baseline, Week 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up. Use the following parameters: Pulse, Temprature and Respiration Rate (3 parameters).

Table 14.3-4.1 Change from Baseline in ECG Values (Safety Analysis Set)

See table 14.3-2.1 for layout. Use footnote below.

Note: Baseline is defined as the last available assessment on or prior to the first dose of study medication. Source Data: Listing 16.2-10.2

Programming note: use timepoints of Baseline, Week 24, 60, 96, 97 and 1 week follow-up.

Table 14.3-4.2

Overall ECG Interpretations and Abnormal Findings (Safety Analysis Set)

| Visit | EGT0001442 | Placebo |
|----------------------------|-------------|-------------|
| Assessment | (N=xxx) | (N=xxx) |
| Screening | | |
| n | xxx | xxx |
| Normal | xxx (xx.x%) | xxx (xx.x%) |
| Abormal | xxx (xx.x%) | xxx (xx.x%) |
| Clinically Significant | xxx (xx.x%) | xxx (xx.x%) |
| Not Clinically Significant | xxx (xx.x%) | xxx (xx.x%) |
| Missing | xxx (xx.x%) | xxx (xx.x%) |
| Week 0 | | |
| n | xxx | xxx |
| Normal | xxx (xx.x%) | xxx (xx.x%) |
| Abormal | xxx (xx.x%) | xxx (xx.x%) |
| Clinically Significant | xxx (xx.x%) | xxx (xx.x%) |
| Not Clinically Significant | xxx (xx.x%) | xxx (xx.x%) |
| Missing | xxx (xx.x%) | xxx (xx.x%) |

Source Data: Listing 16.2-10.3

Programming note: use all available timepoints per data following order such as Screening, Week 0, 24, 60, 96, 97 and 1 week follow-up.

Table 14.3-4.3
ECG Results by Category and Visit
(Safety Analysis Set)

| Parameter<br>Visit | | 0001442<br>=xxx) | | acebo |
|------------------------------|------|------------------|-----|---------|
| ATRIC | ( IN | =xxx) | (IV | (=xxx) |
| QT Range (msec) | | | | |
| Week -5 | | | | |
| n | | xxx | | xxx |
| < 450 | xxx | (xx.x%) | xxx | (xx.x%) |
| >= 450 - < 480 | xxx | (xx.x%) | xxx | (xx.x%) |
| >= 480 - < 500 | xxx | (xx.x%) | xxx | (xx.x%) |
| >= 500 | xxx | (xx.x%) | xxx | (xx.x%) |
| Week 0 | | | | |
| n | | xxx | | xxx |
| < 450 | ~~~ | (xx.x%) | | (xx.x%) |
| >= 450 - < 480 | | (xx.x%) | | (xx.x%) |
| >= 480 - < 500 | | (xx.x%) | | (xx.x%) |
| >= 500 | | (xx.x%) | | (xx.x%) |
| >= 300 | AAA | (22.20) | AAA | (AA:AO) |
| QTcB Range (msec) | | | | |
| Week -5 | | | | |
| n | | xxx | | xxx |
| < 450 | xxx | (xx.x%) | xxx | (xx.x%) |
| >= 450 - < 480 | xxx | (xx.x%) | xxx | (xx.x%) |
| >= 480 - < 500 | xxx | (xx.x%) | xxx | (xx.x%) |
| >= 500 | xxx | (xx.x%) | xxx | (xx.x%) |
| Office Bongo (mang) | | | | |
| QTcF Range (msec)<br>Week -5 | | | | |
| n | | xxx | | xxx |
| < 450 | *** | (xx.x%) | | (xx.x%) |
| >= 450 - < 480 | | (xx.x%) | | (xx.x%) |
| >= 480 - < 500 | | (xx.x%) | | (xx.x%) |
| >= 500 | | | | |
| >= 500 | XXX | (xx.x%) | XXX | (xx.x%) |

Source Data: Listing 16.2-10.2

Programming Note: use all available timepoints per data following order such as Week -5, 0, 24, 60, 96, 97 and 1 week follow-up.

Table 14.3-5.1 Physical Examination (Safety Analysis Set)

| EGT0001442<br>(N=xxx) | Placebo<br>(N=xxx) |
|---|---|
| xxx | xxx |
| xxx (xx.x%) | xxx (xx.x%) |
| xxx (xx.x%) | xxx (xx.x%) |
| xxx (xx.x%) | xxx (xx.x%) |
| xxx | XXX |
| xxx (xx.x%) | xxx (xx.x%) |
| xxx (xx.x%) | xxx (xx.x%) |
| xxx (xx.x%) | xxx (xx.x%) |
| xxx | xxx |
| xxx (xx.x%) | xxx (xx.x%) |
| xxx (xx.x%) | xxx (xx.x%) |
| | XXX XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) XXX XXX (XX.X%) XXX XXX (XX.X%) XXX (XX.X%) XXX (XX.X%) |

Source Data: Listing 16.2-10.4

Programming note: use timepoints of Screening, Week 0, 2, 6, 12, 18, 24, 36, 48, 60, 72, 84, 96, 97 and 1 week follow-up. Complete physical exam is done at Screening, Week 12, 24, 48, 72, 96, 97 and 1 week follow-up. Brief physical exam is done at all other visits. Use all available timepoints per data following order above.

Protocol: THR-1442-C-418 Page x of y

Table 14.3-6.1 NMP22 Test Results (Safety Analysis Set)

| xxx | xxx |
|-------------|-------------|
| xxx (xx.x%) | xxx (xx.x%) |
| xxx (xx.x%) | xxx (xx.x%) |
| | xxx (xx.x%) |

Source Data: Listing 16.2-10.6

Programming note: use all available timepoints per data.

Protocol: THR-1442-C-418 Page x of y

Listing 14.3-1.1
Deaths
(Safety Analysis Set)

Treatment: EGT0001442

| Subject ID/<br>Age/ Sex/ Race [1] | Preferred Term/<br>Vertatim Text | Treatment<br>Emergent<br>Flag | Onset Date/<br>Date of<br>Resolution | Severity/<br>Outcome | Serious/<br>Withdrawn? | Action Taken/<br>Related to<br>Study Drug? |
|---|---|---|---|---|---|---|
| XXXXXX/ | DROWNING/ | Y | 2009-07-25/ | SEVERE/ | YES/ | STUDY DRUG |
| XX/ X/ X | ACCIDENTAL DROWNING | | 2009-07-25 | DEATH DUE TO AE | YES | DISCONTINURED/<br>NO |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Programming Note: Present EGT0001442, and then Placebo treatment groups with each treatment group starting on a new page.

Protocol: THR-1442-C-418 Page x of y

Listing 14.3-2.1 Serious Non-fatal Adverse Events (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Listing 14.3-3.1

Adverse Events Leading to Treatment Discontinuation (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 14.3-4.1 Cardiovascular Adverse Events (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Listing 14.3-5.1 Hypoglycemic Adverse Event (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

## Listing 14.3-6.1 Severe Hypoglycemic Adverse Events (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Listing 14.3-7.1
Renal and Urinary Adverse Events
(Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

## Listing 14.3-8.1 Genitourinary Adverse Events (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Listing 14.3-9.1 Liver Adverse Events (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.
Protocol: THR-1442-C-418 Page x of y

Listing 14.3-10.1 Cancer Adverse Events (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Listing 14.3-11.1 Bone Fracture Adverse Events (Safety Analysis Set)

See Listing 14.3-1.1 for layout. Use footnotes below.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 14.3-12.1

Clinically Significant Abnormal Hematology Laboratory Evaluations

(Safety Analysis Set)

| Subject ID/<br>Age/ Sex/ Race<br>[1] | Visit | Assessment<br>Date | Study<br>Day | Analysis<br>Visit | Lab Test | Value<br>(Unit) | Normal Range |
|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxxx | xxx | xxx | xxx | xxx | xxx (xx) | xxx - xxx |
| 1111, 11, 11 | xxxx | xxx | xxx | xxx | xxx | xxx (xx) | xxx - xxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

### Listing 14.3-12.2 Clinically Significant Abnormal Chemistry Laboratory Evaluations (Safety Analysis Set)

See listing 14.3-12.1 for layout. Use the following footnote.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Listing 14.3-12.3 Clinically Significant Abnormal Urinalysis Laboratory Evaluations (Safety Analysis Set)

See listing 14.3-12.1 for layout. Use the following footnote.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

## Listing 16.1-1.1 Randomized Allocation to Treatment (All Randomized Subjects)

| Subject ID/<br>Age/ Sex/ Race [1] | Randomization Number | Treatment Number | Treatment Description |
|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxxxx | xxx | xxxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-1.1 Subject Disposition (All Randomized Subjects)

| Subject ID/<br>Age/ Sex/ Race [1] | Informed<br>ConsentDate/<br>Randomization<br>Date | Date of<br>First Dose/<br>Last Dose | Date of Last<br>Visit | Study Completion/<br>Reason (if no) | Unblinded during<br>the Study/Date &<br>Reason (if yes) |
|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxxxx/<br>xxxxx | xxxx/<br>xxxx | xxxx | xxx | xxxxxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

## Listing 16.2-2.1 Inclusion/Exclusion Criteria Not Met (All Run-in Failures)

| Subject ID/<br>Age/ Sex/ Race [1] | Protocol<br>Version Date | Criterion Number | Criterion Description |
|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | yyyy-mm-dd | IN01 | xxxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

<DIRECTORY PATH>PROGRAM NAME Executed: DDMMMYYYY hh:mm Data Extracted: DDMONYYYY

Final - 22November2011 

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-2.2
Protocol Deviations
(All Randomized Subjects)

| Subject ID/ | Visit/ | |
|--------------------|------------|--------------------|
| Age/ Sex/ Race [1] | Visit Date | Protocol Deviation |
| XXXXXX/ | Week 12/ | xxxxxxxx |
| XX/ X/ X | | |
| | yyyy-mm-dd | |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-2.3
Major Protocol Deviations
(All Randomized Subjects)

Treatment: EGT0001442

Subject ID/

Age/ Sex/ Race [1] Major Protocol Deviation

XXXXXX/ XX/ X/ X xxxxxxxxxxxxxxxxxxxxx

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-3.1
Analysis Populations
(All Randomized Subjects)

| Subject ID/<br>Age/ Sex/ Race [1] | Randomized | Full Analysis Set | Safety Analysis Set | Per Protocol Analysis Set |
|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | Yes | Yes | Yes | No |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-4.1 Demographic Characteristics (Safety Analysis Set)

| Subject ID/ | | | | | Child | | | |
|---|---|---|---|---|---|---|---|---|
| Age/ Sex/<br>Race [1] | Country/<br>Site | Date of<br>Birth | Race | Ethnicity | Bearing<br>Potential | Height<br>(cm) | Body Mass Index (BMI) (kg/m²) | Baseline HbAlc<br>Category |
| XXXXXX/<br>XX/ X/ X | xxx | xxx | OTHER: xxx | xxx | xxx | xxx | xxx | xxxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-4.2 Substance Use (Safety Analysis Set)

| Subject ID/<br>Age/ Sex/ Race [1] | Screening Visit<br>Date | Consume Alcohol?/<br>If Yes, Units per<br>Week | Tobacco Use?/If<br>Available, Last<br>Tobacco Use Date | Drug Dependecy?/<br>If Yes, Detail/<br>Last Drug Use Date |
|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxxxx | xxxxx | xxxx/xxx | xxxxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-4.3 Drug Screen Results (Safety Analysis Set)

Treatment: EGT0001442

| Subject ID/<br>Age/ Sex/ Race [1] | Assessment Date | Parameter | Result (unit) |
|---|---|---|---|
| Age/ Sex/ Race [1] | Assessment Date | Parameter | Result (unit) |
| XXXXXX/<br>XX/ X/ X | xxxxx | HBsAG | Negative |
| . , | | HBcAG | Negative |
| | | HCV Ab | xxx |
| | | Amphetamines | xxx |
| | | Barbiturates | xxx |
| | | Cocaine | xxx |
| | | Metabolites | XXX |
| | | Opiates | XXX |
| | | Benzodiazepines | XXX |
| | | Cannabinoids | XXX |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-4.4 Medical History (Safety Analysis Set)

| Subject ID/ | | | |
|--------------------|-----------|------------|----------|
| Age/ Sex/ Race [1] | Condition | Start Date | End Date |
| XXXXXX/ | XXXXX | xxxxx | xxxxxx |
| XX/ X/ X | | | |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418

Listing 16.2-4.5 Diabetes Medical History (Safety Analysis Set) Page x of y

| Subject ID/<br>Age/ Sex/ Race [1] | Condition | Assessment | Result |
|-----------------------------------|-----------|---------------|--------|
| XXXXXX/ | Blindness | Eye Affected | Left |
| XX/ X/ X | | Date of Onset | xxxxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-5.1
Prior and Concomitant Medications
(Safety Analysis Set)

Treatment: EGT0001442

| Subject ID/<br>Age/ Sex/ Race<br>[1] | Preferred Term/<br>Vertatim Text | Med. Type | Dose/<br>Units/<br>Freq/<br>Route | Date<br>Started/<br>Date<br>Stopped | Indication | Anti-<br>diabetic<br>Med? | Rescue<br>Med? | Used to<br>Treat an AE? |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | ATENOLOL/<br>ATENOLOL | Prior, Cor | 50/<br>MILLIGRAM/<br>ONCE DAILY/<br>ORAL | 2007/xxxx | xxxxxx | Yes | Yes | Yes |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

<sup>[2]</sup> Prior=Prior medication, Con=Concomitant medication.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-6.1 Study Drug Administration (Safety Analysis Set)

| Subject ID/<br>Age/ Sex/ Race [1] | Visit | Dispensed?/If No,<br>Reason | Dispense<br>Date | # of<br>Capsules<br>Dispensed | Kit(s)<br>Dispensed | # of<br>Capsules<br>Returned | Kit(s)<br>Returned |
|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxx | xxx | xxx | xxx | xxx | xxx | xxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-7.1 HbA1c (%) (Full Analysis Set)

| Subject ID/<br>Age/ Sex/ Race [1] | Visit | Assessment<br>Date | Study Day | Analysis<br>Visit | Post-<br>rescue? | Value | Baseline<br>[2] | Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxx | xxx | xxx | xxx | No | xxx | xxx | xxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

<sup>[2]</sup> Baseline is defined as the last available assessment on or prior to the first dose of study medication.

Protocol: THR-1442-C-418 Page x of y

## Listing 16.2-7.2 Fasting Plasma Glucose (mmol/L) (Full Analysis Set)

#### See Listing 16.2-7.1 for layout. Use footnotes below.

- [1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.
- [2] Baseline is defined as the last available assessment on or prior to the first dose of study medication.

Listing 16.2-7.3
Weight(kg)
(Full Analysis Set)

#### See Listing 16.2-7.1 for layout. Use footnotes below.

- [1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.
- [2] Baseline is defined as the last available assessment on or prior to the first dose of study medication.

Protocol: THR-1442-C-418 Page x of y

## Listing 16.2-7.4 Systolic Blood Pressure (mmHg) (Full Analysis Set)

| Subject ID/<br>Age/ Sex/<br>Race [1] | Visit | Assessment<br>Date | Study Day | Analysis<br>Visit | Post-<br>rescue? | 1 <sup>st</sup> /<br>2 <sup>nd</sup><br>Measure | Mean of 2<br>Measures | Baseline<br>[2] | Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxx | xxx | xxx | xxx | No | xxxx | xxx | xxx | xxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

<sup>[2]</sup> Baseline is defined as the last available assessment on or prior to the first dose of study medication.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-7.5
Diastolic Blood Pressure (mmHg)
(Full Analysis Set)

See Listing 16.2-7.4 for layout. Use footnotes below.

- [1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.
- [2] Baseline is defined as the last available assessment on or prior to the first dose of study medication.

Listing 16.2-8.1 Adverse Events (Safety Analysis Set)

See Listing 14.3-1.1 for layout.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418

### Listing 16.2-8.2 Hypoglycemic Events Supplemental Information (Safety Analysis Set)

Page x of y

| Subject ID/<br>Age/ Sex/ Race [1] | Preferred Term/<br>Vertatim Text | Treatment<br>Emergent<br>Flag | Onset Date/<br>Date of<br>Resolution | ADA Severity | Intervention |
|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | DROWNING/<br>ACCIDENTAL<br>DROWNING | Y | 2009-07-25/<br>2009-07-25 | xxxxxxx | xxxxxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

### Listing 16.2-9.1 Hematology Laboratory Evaluations (Safety Analysis Set)

Treatment: EGT0001442

| Subject ID/ | | | | | | | | | Flag [2] |
|---|---|---|---|---|---|---|---|---|---|
| Age/ Sex/ Race<br>[1] | Visit | Assessment<br>Date | Study<br>Day | Analysis<br>Visit | Lab Test | Value<br>(Unit) | Normal Range | NR | CS |
| XXXXXX/<br>XX/ X/ X | xxxx | xxx | xxx | xxx | xxx | xxx (xx) | xxx - xxx | xx | xx |
| AA/ A/ A | xxxx | xxx | xxx | xxx | xxx | xxx (xx) | xxx - xxx | xx | xx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

<sup>[2]</sup> NR for Normal Range flag, CS for Clinical Significance flag. H=Above range, L=Below range. CS=Clinically significant, NCS=Not clinically significant.

Protocol: THR-1442-C-418 Page x of y

### Listing 16.2-9.2 Chemistry Laboratory Evaluations (Safety Analysis Set)

#### See listing 16.2-9.1 for layout. Use the following footnote.

- [1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.
- [2] NR for Normal Range flag, CS for Clinical Significance flag. H=Above range, L=Below range. CS=Clinically significant, NCS=Not clinically significant.

Listing 16.2-9.3
Urinalysis Laboratory Evaluations
(Safety Analysis Set)

#### See listing 16.2-9.1 for layout. Use the following footnote.

- [1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.
- [2] NR for Normal Range flag, CS for Clinical Significance flag. H=Above range, L=Below range. CS=Clinically significant, NCS=Not clinically significant.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-10.1 Vital Signs (Safety Analysis Set)

Treatment: EGT0001442

| Subject ID/<br>Age/ Sex/ Race [1] | Visit | Assessment Date | Study Day | Analysis Visit | Parameter | Result (Unit) |
|---|---|---|---|---|---|---|
| XXXXXX/ | xxx | xxxx | xx | xxx | xx | xx (xx) |
| XX/ X/ X | | | | | | |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Programming note: use the following parameters: Pulse, Temprature and Respiration Rate (3 parameters).

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-10.2 ECG Values (Safety Analysis Set)

See listing 16.2-10.1 for layout. Use the following footnote.

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418

# Listing 16.2-10.3 Overall ECG Interpretations and Abnormal Findings (Safety Analysis Set)

Page x of y

Treatment: EGT0001442

| Subject ID/<br>Age/ Sex/ Race [1] | Visit | Assessment<br>Date | Study Day | Analysis<br>Visit | Overall<br>Interpretation | Abnormal<br>Findings | CS Flag [2] |
|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxx | xxxx | xx | xxx | Abnormal | xxx | xxx |
| M $M$ $M$ | xxx | xxxx | xx | xxx | xxx | xxx | |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

<sup>[2]</sup> CS flag for Clinical Significance flag. CS=Clinically significant, NCS=Not clinically significant.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-10.4 Physical Examinations (Safety Analysis Set)

| Subject ID/<br>Age/ Sex/ Race [1] | Visit | Assessment<br>Date | Study Day | Analysis<br>Visit | Assessment | Status | Specify if<br>Abnormality |
|---|---|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxx | xxxx | xx | xxx | xxx | Normal | |
| AA/ A/ A | xxx | xxxx | xx | xxx | xxx | Abnormal | xxx |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-10.5 Pregnancies (Safety Analysis Set)

Treatment: EGT0001442

Subject ID/ Age/ Sex/ Race [1]

XXXXXX/ XX/ X/ X

[1] Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.

Programming note: Display only 'There are no observations to this table.' If no events.

Protocol: THR-1442-C-418 Page x of y

Listing 16.2-10.6 NMP22 Testing Results (Safety Analysis Set)

Treatment: EGT0001442

| Subject ID/<br>Age/ Sex/ Race [1] | Visit | Assessment<br>Date | Study Day | Assessment | If Positive, Urine<br>Culture?/Culture Result | Investigator<br>Comment |
|---|---|---|---|---|---|---|
| XXXXXX/<br>XX/ X/ X | xxx | xxxx | xx | Positive | Yes/xxxxx | xxx |
| 1111, 11, 11 | xxx | xxxx | xxx | Negative | | |
| | AAA | XXXX | AAA | Negacive | | |

<sup>[1]</sup> Sex: F=Female, M=Male; Race: W=White, B=Black, A=Asian, I=American Indian or Alaska Native, H=Native Hawaiian or Other Pacific Islander, O=Other.